CLINICAL TRIAL: NCT03732807
Title: A PHASE 2B/3 RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, DOSE-RANGING STUDY TO INVESTIGATE THE EFFICACY AND SAFETY OF PF-06651600 IN ADULT AND ADOLESCENT ALOPECIA AREATA (AA) SUBJECTS WITH 50% OR GREATER SCALP HAIR LOSS
Brief Title: PF-06651600 for the Treatment of Alopecia Areata
Acronym: ALLEGRO-2b/3
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7981015; 2018-001714-14 (EudraCT Number); ALLEGRO 2B/3 (Other: Alias Study Number)
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Results first posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Alopecia Areata
Keywords: Alopecia; Alopecia totalis; Alopecia universalis; Patchy hair loss; Diffuse hair loss; Hair loss; Hair disease; PF-06651600; Ritlecitinib
MeSH Terms: conditions — Alopecia Areata; Alopecia; Alopecia universalis; Hair Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Sequence A (Experimental): Induction dose given once daily (QD) for 4 weeks followed by maintenance dose #1 given QD for 44 weeks
  Interventions: Drug: PF-06651600 Induction Dose; Drug: PF-06651600 Maintenance Dose #1
- Sequence B (Experimental): Induction dose given QD for 4 weeks followed by maintenance dose #2 given QD for 44 weeks
  Interventions: Drug: PF-06651600 Induction Dose; Drug: PF-06651600 Maintenance Dose #2
- Sequence C (Experimental): Maintenance dose #1 given QD for 48 weeks
  Interventions: Drug: PF-06651600 Maintenance Dose #1
- Sequence D (Experimental): Maintenance dose #2 given QD for 48 weeks
  Interventions: Drug: PF-06651600 Maintenance Dose #2
- Sequence E (Experimental): Maintenance dose #3 given QD for 48 weeks
  Interventions: Drug: PF-06651600 Maintenance Dose #3
- Sequence F (Experimental): Placebo given QD for 24 weeks followed by induction dose given QD for 4 weeks then maintenance dose #1 given QD for 20 weeks
  Interventions: Drug: PF-06651600 Induction Dose; Drug: PF-06651600 Maintenance Dose #1; Drug: Placebo
- Sequence G (Experimental): Placebo given QD for 24 weeks followed by maintenance dose #1 given QD for 24 weeks
  Interventions: Drug: PF-06651600 Maintenance Dose #1; Drug: Placebo

INTERVENTIONS:
Drug: PF-06651600 Induction Dose — Oral tablets taken once daily (QD)
  Arms: Sequence A; Sequence B; Sequence F
Drug: PF-06651600 Maintenance Dose #1 — Oral tablets taken QD
  Arms: Sequence A; Sequence C; Sequence F; Sequence G
Drug: PF-06651600 Maintenance Dose #2 — Oral tablets taken QD
  Arms: Sequence B; Sequence D
Drug: PF-06651600 Maintenance Dose #3 — Oral tablets taken QD
  Arms: Sequence E
Drug: Placebo — Oral tablets taken QD
  Arms: Sequence F; Sequence G

SUMMARY:
This is a global Phase 2b/3 study to evaluate the safety and effectiveness of an investigational study drug (called PF-06651600) in adults and adolescents (12 years and older) who have 50% or greater scalp hair loss. The study is placebo-controlled, meaning that some patients entering the study will not receive active study drug but will receive tablets with no active ingredients (a placebo). This is a dose-ranging study, investigating 5 different dosing regimens. It will be double-blinded, meaning that the sponsor, the study doctors, the staff, and the patients will not know whether a patient is on active study drug (or the dose) or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of alopecia areata with no other cause of hair loss
* ≥50% hair loss of the scalp, including alopecia totalis and alopecia universalis, without evidence of terminal hair regrowth within 6 months
* Current episode of hair loss ≤10 years

Exclusion Criteria:

* Other types of alopecia or other diseases that can cause hair loss
* Other scalp diseases that could interfere with assessment of hair loss/regrowth
* Subjects with shaved heads must not enter the study until hair has grown back & is considered stable by the investigator
* Any previous use of any Janus kinase (JAK) inhibitor

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 718 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (154):
- United States (45):
  - The University of Alabama at Birmingham Hospital Outreach Lab, Birmingham, Alabama
  - The University of Alabama at Birmingham, Department of Dermatology, Birmingham, Alabama
  - Mosaic Dermatology, Beverly Hills, California
  - University of California, Irvine, Department of Dermatology, Dermatology Clinical Research Center, Irvine, California
  - Dermatology Specialists, Inc., Murrieta, California
  - University of California, San Francisco, San Francisco, California
  - Kaiser Permanente Clinical Trials Unit, San Francisco, California
  - Southern California Dermatology, Inc., Santa Ana, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Colorado Hospital Clinical and Translational Research Center, Aurora, Colorado
  - University of Colorado Hospital Outpatient Pavillion, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Church Street Research Unit, New Haven, Connecticut
  - Medstar Georgetown University Hospital Center-Department of Otolaryngology, Washington D.C., District of Columbia
  - Medstar Washington Hospital Center-Claude Nogay Research Pharmacy, Washington D.C., District of Columbia
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Medstar Georgetown University Hospital Center-Department of Pediatrics, Washington D.C., District of Columbia
  - Siperstein Dermatology Group, Boynton Beach, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Advanced Clinical Research, Meridian, Idaho
  - Northwestern Medical Group, Chicago, Illinois
  - Northwestern Medicine Diagnostic Testing Center, Chicago, Illinois
  - Northwestern Medicine, Chicago, Illinois
  - Northwestern Memorial Hospital, Investigational Research Pharmacy, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - NorthShore University HealthSystem, Skokie, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics; Department of Pharmacy-IDS;, Iowa City, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Medstar Georgetown University Hospital - Department of Dermatology, Chevy Chase, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota Department of Dermatology, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Investigational Drug Services Attn: Darlette Luke, Minneapolis, Minnesota
  - Skin Specialists, PC, Omaha, Nebraska
  - The Dermatology Group, P.C., Verona, New Jersey
  - NYU School of Medicine, The Ronald O. Perelman Department of Dermatology, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - UNC CTRC, Chapel Hill, North Carolina
  - UNC Hospitals, Investigational Drug Service, Chapel Hill, North Carolina
  - UNC Dermatology Clinical Trials Unit, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Vital Prospects Clinical Research Institute, P.C, Tulsa, Oklahoma
  - The University of Texas Health Science Center at Houston, Houston, Texas
- Argentina (2):
  - CINME Centro de Investigaciones Metabolicas, CABA, Buenos Aires
  - Psoriahue Medicina Interdisciplinaria, CABA
- Australia (8):
  - Premier Specialists Pty Ltd, Kogarah, New South Wales
  - St George Dermatology and Skin Cancer Centre, Kogarah, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
  - Skin Health Institute, Carlton, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Royal Park Campus, Parkville, Victoria
- Canada (12):
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Eastern Canada Cutaneous Research Associates Ltd., Halifax, Nova Scotia
  - Medicor Research Inc, Greater Sudbury, Ontario
  - Sudbury Skin Clinique, Greater Sudbury, Ontario
  - Guenther Research Inc, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - The Centre for Clinical Trials, Oakville, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - York Dermatology Clinic and Research Centre, Richmond Hill, Ontario
  - Research Toronto, Toronto, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec metropolitain, Québec, Quebec
- Chile (4):
  - Centro Internacional de Estudios Clinicos, CIEC, Santiago, Recoleta
  - Medical Skin Center, Viña del Mar, Región de Valparaíso
  - Centro Medico Skin Med, Santiago, Santiago Metropolitan
  - Clinica Dermacross S.A., Santiago, Santiago Metropolitan
- China (11):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen, Guangdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Huashan Hospital, Fudan University/Dermatology Department, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of College of Medicine, Zhejiang University/Dermatology Dept, Hangzhou, Zhejiang
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai
- Colombia (3):
  - Fundacion Centro de Investigacion Clinica CIC, Medellín, Antioquia
  - Fundacion Hospitalaria San Vicente de Paul, Medellín, Antioquia
  - Centro de Investigación en Reumatología y Especialidades Médicas SAS - CIREEM SAS, Bogotá, D.C.
- Czechia (5):
  - DERMAMEDICA s.r.o., Náchod
  - Fakultni nemocnice Olomouc, Olomouc
  - Clintrial s.r.o., Prague
  - Sanatorium profesora Arenbergera, Prague
  - Nemocnice Na Bulovce, Praha 8- Liben
- Germany (6):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Emovis GmbH, Berlin
  - Universitaetsklinikum Erlangen, Erlangen
  - University Hospital Frankfurt, Frankfurt am Main
  - University Hospital Schleswig-Holstein, Lübeck
  - University Hospital Muenster, Münster
- Hungary (4):
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem, Debrecen
  - Bugat Pal Korhaz, Borgyogyaszat, Gyöngyös
  - Szegedi Tudományegyetem Altalanos Orvostudomanyi Kar, Szeged
- Japan (6):
  - Nagoya City University Hospital - Dermatology, Nagoya, Aichi-ken
  - Tohoku University hospital, Sendai, Miyagi
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Juntendo Tokyo Koto Geriatric Medical Center, Koto-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Osaka City University Hospital, Osaka
- Mexico (2):
  - Sociedad de Metabolismo y Corazon S.C., Veracruz
  - Hospital D'Maria, Veracruz
- Poland (8):
  - Centermed Krakow Sp.z o.o., Krakow
  - Medicover Sp.z.o.o, Lodz
  - Dermoklinika Centrum Medyczne s.c., M. Kierstan, J. Narbutt, A. Lesiak, Lodz
  - Sanova Audiological Care Polska Sp.z.o.o, Lodz
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - RCMed Oddzial Warszawa, Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
  - Cityclinic Przychodnia Lekarsko Psychologiczna Matusiak Spółka Partnerska, Wroclaw
- Russia (9):
  - State Budgetary Healthcare Institution Chelyabinsk Regional Clinical Dermatovenerologic Dispensary, Chelyabinsk
  - University Clinic of Kirov SMU, Kirov
  - Clinical Medical Center of A.I. Yevdokimov MSMSU, Moscow
  - Federal State Autonomous Institution National Medical Research Centre of Childrens Health, Moscow
  - State Budgetary Institution of the Rostov Region "Dermatovenerologic Dispensary", Rostov-on-Don
  - Limited Liability Company "Centre Vitiligo" ("Centre Vitiligo" LLC), Saint Petersburg
  - Limited Liability Company "Pierre Volkenshtein Skin Diseases Clinic", Saint Petersburg
  - Saint Petersburg State Budgetary Healthcare Institution "Dermatovenerologic Dispensary No. 10 -, Saint Petersburg
  - State Autonomous Healthcare Institution of the Yaroslavl Region Clinical Emergency Hospital, Yaroslavl
- South Korea (2):
  - Pusan National University Hospital, Busan
  - Seoul National University Hospital, Seoul
- Spain (10):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Reina Sofía, Servicio Dermatologia, Córdoba
  - Servicio Otorrinolaringologia, Hospital Universitario Reina Sofia, Córdoba
  - Servicio Radiologia, Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Servicio de Dermatologia, Hospital Universitario y Politecnico La Fe, Valencia
  - Servicio de Otorrinolaringologia, Hospital Universitario y Politecnico La Fe, Valencia
  - Servicio de Radiologia, Hospital Universitario y Politecnico Le Fe, Valencia
- Taiwan (7):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - CHANG GUNG MEMORIAL HOSPITAL Kaohsiung Branch, Kaohsiung City
  - Taipei Medical University-Shuang Ho Hospital, Ministry of Health and Welfare, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - Chung-Shan Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital-Linkou Branch, Taoyuan
- United Kingdom (10):
  - Brighton and Sussex University Hospitals NHS Trust, Brighton, EAST Sussex
  - Southampton University Hospital NHS Foundation Trust, Royal South Hants Hospital, Southampton, Hampshire
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - NHS Tayside Ninewells Hospital, Dundee
  - NHS Greater Glasgow and Clyde Queen Elizabeth University Hospital, Glasgow
  - NHS Greater Glasgow and Clyde, Glasgow
  - Southampton University Hospital NHS Foundation Trust, University Hospital Southampton, Hampshire
  - Harley Grove Medical Centre, London
  - Guy's and St.Thomas' Hospitals NHS Foundation Trust, St.Thomas' Hospital,, London
  - Guy's and St.Thomas' Hospitals NHS Foundation Trust, Guy's Hospital,, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Mostaghimi A, Gibson A, Dwyer G, Oluboyede Y, Mazar I, Gorbatenko-Roth K, Law E. Exploring Factors That Influence the Measurement of Patient-Reported Impacts of Alopecia Areata. Dermatol Ther (Heidelb). 2025 Jun;15(6):1391-1403. doi: 10.1007/s13555-025-01400-7. Epub 2025 Apr 22. PMID 40261547
- [Derived] King B, Mirmirani P, Lo Sicco K, Ramot Y, Sinclair R, Asfour L, Ezzedine K, Paul C, Ohyama M, Edwards RA, Bonfanti G, Kerkmann U, Wajsbrot D, Ishowo-Adejumo R, Zwillich SH, Lejeune A. Patterns of clinical response in patients with alopecia areata treated with ritlecitinib in the ALLEGRO clinical development programme. J Eur Acad Dermatol Venereol. 2025 Jun;39(6):1163-1173. doi: 10.1111/jdv.20547. Epub 2025 Feb 17. PMID 39962358
- [Derived] Sinclair R, Mesinkovska N, Mitra D, Wajsbrot D, Law EH, Wolk R, King B. Patient-Reported Hair Loss and Its Impacts as Measured by the Alopecia Areata Patient Priority Outcomes Instrument in Patients Treated with Ritlecitinib: The ALLEGRO Phase 2b/3 Randomized Clinical Trial. Am J Clin Dermatol. 2025 Jan;26(1):109-119. doi: 10.1007/s40257-024-00899-4. Epub 2024 Oct 23. PMID 39441519
- [Derived] Mesinkovska N, King B, Zhang X, Guttman-Yassky E, Magnolo N, Sinclair R, Mizuashi M, Shapiro J, Peeva E, Banerjee A, Takiya L, Cox LA, Wajsbrot D, Kerkmann U, Law E, Wolk R, Schaefer G. Efficacy and safety of ritlecitinib, an oral JAK3/TEC family kinase inhibitor, in adolescent and adult patients with alopecia totalis and alopecia universalis. J Dermatol. 2024 Nov;51(11):1414-1424. doi: 10.1111/1346-8138.17442. Epub 2024 Sep 27. PMID 39328096
- [Derived] Fu J, Egeberg A, Holmes S, Vano-Galvan S, Steinhoff M, Edwards R, Bonfanti G, Nagra R, Wolk R, Tran H, Law E. Impact of Previous Alopecia Areata Treatment on Efficacy Responses up to Week 48 Following Ritlecitinib Treatment: A Post Hoc Analysis. Dermatol Ther (Heidelb). 2024 Oct;14(10):2759-2769. doi: 10.1007/s13555-024-01260-7. Epub 2024 Sep 10. PMID 39254890
- [Derived] King B, Soung J, Tziotzios C, Rudnicka L, Joly P, Gooderham M, Sinclair R, Mesinkovska NA, Paul C, Gong Y, Anway SD, Tran H, Wolk R, Zwillich SH, Lejeune A. Integrated Safety Analysis of Ritlecitinib, an Oral JAK3/TEC Family Kinase Inhibitor, for the Treatment of Alopecia Areata from the ALLEGRO Clinical Trial Program. Am J Clin Dermatol. 2024 Mar;25(2):299-314. doi: 10.1007/s40257-024-00846-3. Epub 2024 Jan 23. PMID 38263353
- [Derived] Wojciechowski J, S Purohit V, Huh Y, Banfield C, Nicholas T. Evolution of Ritlecitinib Population Pharmacokinetic Models During Clinical Drug Development. Clin Pharmacokinet. 2023 Dec;62(12):1765-1779. doi: 10.1007/s40262-023-01318-3. Epub 2023 Nov 2. PMID 37917289
- [Derived] Thaci D, Tziotzios C, Ito T, Ko J, Karadag AS, Fang H, Edwards RA, Bonfanti G, Wolk R, Tran H, Law E. Hair Loss Profiles and Ritlecitinib Efficacy in Patients with Alopecia Areata: Post Hoc Analysis of the ALLEGRO Phase 2b/3 Study. Dermatol Ther (Heidelb). 2023 Nov;13(11):2621-2634. doi: 10.1007/s13555-023-00997-x. Epub 2023 Sep 14. PMID 37707764
- [Derived] King B, Zhang X, Harcha WG, Szepietowski JC, Shapiro J, Lynde C, Mesinkovska NA, Zwillich SH, Napatalung L, Wajsbrot D, Fayyad R, Freyman A, Mitra D, Purohit V, Sinclair R, Wolk R. A plain language summary on ritlecitinib treatment for adults and adolescents with alopecia areata. Immunotherapy. 2023 Oct;15(14):1093-1103. doi: 10.2217/imt-2023-0069. Epub 2023 Jul 5. PMID 37403610
- [Derived] King B, Zhang X, Harcha WG, Szepietowski JC, Shapiro J, Lynde C, Mesinkovska NA, Zwillich SH, Napatalung L, Wajsbrot D, Fayyad R, Freyman A, Mitra D, Purohit V, Sinclair R, Wolk R. Efficacy and safety of ritlecitinib in adults and adolescents with alopecia areata: a randomised, double-blind, multicentre, phase 2b-3 trial. Lancet. 2023 May 6;401(10387):1518-1529. doi: 10.1016/S0140-6736(23)00222-2. Epub 2023 Apr 14. PMID 37062298
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981015

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 1097 participants signed the informed consent form. Out of which 379 participants were screen failures, 718 actually enrolled into the study and were assigned to study treatments.
Groups:
- Ritlecitinib (PF-06651600) 200 mg Then 50 mg: Participants aged 12 years or above with moderate to severe alopecia areata (AA) with greater than or equal to (>=) 50% hair loss of the scalp were randomized to receive Ritlecitinib 4 of 50 milligram (mg) tablet once daily for 4 weeks (loading phase) and then 50 mg tablet once daily for next 20 weeks (maintenance phase). Participants then entered into extension phase of 24 weeks and continued to receive 50 mg tablet once daily. Participants were followed up to maximum of 5 weeks after the last dose of study drug .
- Ritlecitinib (PF-06651600) 200 mg Then 30 mg: Participants aged 12 years or above with moderate to severe AA with >=50% hair loss of the scalp were randomized to receive Ritlecitinib 4 of 50 mg tablet once daily for 4 weeks (loading phase) and then 3 of 10 mg tablet once daily for next 20 weeks (maintenance phase). Participants then entered into extension phase of 24 weeks and continued to receive 3 of 10 mg tablet once daily. Participants were followed up to maximum of 5 weeks after the last dose of study drug.
- Ritlecitinib (PF-06651600) 50 mg: Participants aged 12 years or above with moderate to severe AA with >=50% hair loss of the scalp were randomized to receive Ritlecitinib 50 mg tablet once daily for 4 weeks (loading phase). Participants then continued to receive 50 mg tablet once daily in maintenance phase of 20 weeks and extension phase of 24 weeks. Participants were followed up to maximum of 5 weeks after the last dose of study drug.
- Ritlecitinib (PF-06651600) 30 mg: Participants aged 12 years or above with moderate to severe AA with >=50% hair loss of the scalp were randomized to receive Ritlecitinib 3 of 10 mg tablet once daily for 4 weeks (loading phase). Participants then continued to receive 3 of 10 mg tablet once daily in maintenance phase of 20 weeks and extension phase of 24 weeks. Participants were followed up to maximum of 5 weeks after the last dose of study drug.
- Ritlecitinib (PF-06651600) 10 mg: Participants aged 12 years or above with moderate to severe AA with >=50% hair loss of the scalp were randomized to receive Ritlecitinib 10 mg tablet once daily for 4 weeks (loading phase). Participants then continued to receive 10 mg tablet once daily in maintenance phase of 20 weeks and extension phase of 24 weeks. Participants were followed up to maximum of 5 weeks after the last dose of study drug.
- Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg: Participants aged 12 years or above with moderate to severe AA with >=50% hair loss of the scalp were randomized to receive placebo once daily for 4 weeks (loading phase) and then continued placebo once daily for next 20 weeks (maintenance phase). Participants then entered into extension phase of 24 weeks and received 4 of 50 mg tablet once daily for 4 weeks and then 50 mg tablet once daily for 20 weeks. Participants were followed up to maximum of 5 weeks after the last dose of study drug.
- Placebo, Ritlecitinib (PF-06651600) 50 mg: Participants aged 12 years or above with moderate to severe AA with >=50% hair loss of the scalp were randomized to receive placebo once daily for 4 weeks (loading phase) and then continued to receive placebo once daily for next 20 weeks (maintenance phase). Participants then entered into extension phase of 24 weeks and received 50 mg tablet once daily. Participants were followed up to maximum of 5 weeks after the last dose of study drug.
Period: Treatment Period (up to Week 24)
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Placebo, Ritlecitinib (PF-06651600) 50 mg
Started | 132 | 130 | 130 | 132 | 63 | 65 | 66
Completed | 122 | 124 | 121 | 117 | 58 | 63 | 61
Not Completed | 10 | 6 | 9 | 15 | 5 | 2 | 5
Not completed — Adverse Event | 3 | 0 | 2 | 4 | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 2 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 2 | 5 | 0 | 0 | 1
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 4 | 4 | 1 | 1 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Treatment Extension (Week 25 up to 48)
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Placebo, Ritlecitinib (PF-06651600) 50 mg
Started | 113 (Participants continued dosing according to their assigned sequence in the preceding period.) | 111 (Participants continued dosing according to their assigned sequence in the preceding period.) | 108 (Participants continued dosing according to their assigned sequence in the preceding period.) | 106 (Participants continued dosing according to their assigned sequence in the preceding period.) | 49 (Participants continued dosing according to their assigned sequence in the preceding period.) | 59 (Participants continued dosing according to their assigned sequence in the preceding period.) | 57 (Participants continued dosing according to their assigned sequence in the preceding period.)
Completed | 107 | 100 | 103 | 97 | 44 | 56 | 53
Not Completed | 6 | 11 | 5 | 9 | 5 | 3 | 4
Not completed — Adverse Event | 0 | 2 | 2 | 1 | 0 | 0 | 2
Not completed — Lack of Efficacy | 2 | 1 | 0 | 3 | 3 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1 | 1 | 2 | 0
Not completed — Non-Compliant with study drug | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 1 | 1 | 0 | 1 | 1
Not completed — Other | 1 | 4 | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized, regardless of whether they received study medication.
Groups:
- Ritlecitinib (PF-06651600) 200 mg Then 50 mg: Participants aged 12 years or above with moderate to severe AA with >=50% hair loss of the scalp were randomized to receive Ritlecitinib 4 of 50 mg tablet once daily for 4 weeks (loading phase) and then 50 mg tablet once daily for next 20 weeks (maintenance phase). Participants then entered into extension phase of 24 weeks and continued to receive 50 mg tablet once daily. Participants were followed up to maximum of 5 weeks after the last dose of study drug .
- Total: Total of all reporting groups
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Placebo, Ritlecitinib (PF-06651600) 50 mg | Total
Number analyzed (Participants) | 132 | 130 | 130 | 132 | 63 | 65 | 66 | 718
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.5 (14.98) | 33.7 (13.75) | 32.4 (13.36) | 33.7 (14.83) | 34.3 (13.88) | 33.0 (14.01) | 35.0 (15.89) | 33.8 (14.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 85 | 71 | 80 | 43 | 46 | 40 | 446
  Male | 51 | 45 | 59 | 52 | 20 | 19 | 26 | 272
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 16 | 11 | 23 | 8 | 7 | 4 | 87
  Not Hispanic or Latino | 113 | 114 | 116 | 109 | 55 | 58 | 61 | 626
  Unknown or Not Reported | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 3
  Asian | 33 | 28 | 43 | 34 | 17 | 14 | 17 | 186
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 6 | 7 | 5 | 3 | 2 | 2 | 2 | 27
  White | 92 | 90 | 79 | 91 | 42 | 47 | 47 | 488
  More than one race | 0 | 3 | 1 | 2 | 0 | 2 | 0 | 8
  Unknown or Not Reported | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Absolute Severity of Alopecia Tool (SALT) Score of Less Than or Equal to 20 at Week 24
Description: SALT is a quantitative assessment of AA severity based on the scalp hair loss. The SALT score can vary from 0 (normal) to 100 (severe), with higher scores representing increased severity of disease. In this outcome measure, percentage of participants with SALT score less than or equal to (<=) 20 at week 24 were reported.
Time Frame: Week 24
Population: FAS included all participants who were randomized, regardless of whether they received study medication. Participants with missing SALT scores due to coronavirus disease-19 related reasons were excluded from this analysis, while participants with missing data due to other reasons were considered as non-responders. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Placebo: Participants aged 12 years or above with moderate to severe AA with>=50% hair loss of the scalp were randomized to receive placebo once daily for 4 weeks (loading phase) and then continued placebo once daily for next 20 weeks (maintenance phase). Participants then entered into extension phase of 24 weeks and received either 4 of 50 mg tablet once daily for 4 weeks followed by 50 mg tablet once daily for next 20 weeks or 50 mg tablet once daily for next 24 weeks. Participants were followed up to maximum of 5 weeks after the last dose of study drug.
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo
Number analyzed (Participants) | 124 | 121 | 124 | 119 | 59 | 130
Percentage of participants | 30.65 [22.53 to 38.76] | 22.31 [14.90 to 29.73] | 23.39 [15.94 to 30.84] | 14.29 [8.00 to 20.57] | 1.69 [0.00 to 4.99] | 1.54 [0.00 to 3.65]
Statistical Analysis 1: Comparison: Ritlecitinib (PF-06651600) 200 mg Then 50 mg vs Placebo; Test type: Superiority; p < 0.000001, Miettinen and Nurminen method; Estimate of difference = 29.11, 95% CI 2-sided [21.17 to 37.91]
Statistical Analysis 2: Comparison: Ritlecitinib (PF-06651600) 200 mg Then 30 mg vs Placebo; Test type: Superiority; p < 0.000001, Miettinen and Nurminen method; Estimate of difference = 20.78, 95% CI 2-sided [13.65 to 29.18]
Statistical Analysis 3: Comparison: Ritlecitinib (PF-06651600) 50 mg vs Placebo; Test type: Superiority; p < 0.000001, Miettinen and Nurminen method; Estimate of difference = 21.85, 95% CI 2-sided [14.65 to 30.23]
Statistical Analysis 4: Comparison: Ritlecitinib (PF-06651600) 30 mg vs Placebo; Test type: Superiority; p = 0.000154, Miettinen and Nurminen method; Estimate of difference = 12.75, 95% CI 2-sided [6.69 to 20.36]

2. Secondary Outcome: Percentage of Participants With an Absolute SALT Score of Less Than or Equal to 10 at Week 24: Analysis 4
Description: SALT is a quantitative assessment of AA severity based on the scalp hair loss. The SALT score can vary from 0 (normal) to 100 (severe), with higher scores representing increased severity of disease. In this outcome measure, percentage of participants with SALT score <= 10 at week 24 were reported.
Time Frame: Week 24
Population: FAS included all participants who were randomized, regardless of whether they received study medication. Analysis 4: Data imputed by using a missing at random (MAR) mechanism for participants with missing data due to COVID-19. Missing data due to reasons not related to COVID-19 were consider as non-responders.
Measure: Number; unit: Percentage of participants
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo
Number analyzed (Participants) | 118 | 119 | 119 | 114 | 55 | 125
Percentage of participants | 21.29 | 12.87 | 13.42 | 10.62 | 1.65 | 1.54
Statistical Analysis 1: Comparison: Ritlecitinib (PF-06651600) 200 mg Then 50 mg vs Placebo; A generalized linear mixed effect model without imputation using observed data up to Week 24 was used as the imputation model. A single complete imputed data set for Week 24 was analyzed using the Miettinen and Nurminen method as the analysis model; Test type: Superiority; p < 0.000001, Miettinen and Nurminen method; Estimate of difference = 19.75, 95% CI 2-sided [11.91 to 27.59]
Statistical Analysis 2: Comparison: Ritlecitinib (PF-06651600) 200 mg Then 30 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.000526, Miettinen and Nurminen method; Estimate of difference = 11.33, 95% CI [4.93 to 17.74]
Statistical Analysis 3: Comparison: Ritlecitinib (PF-06651600) 50 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.000311, Miettinen and Nurminen method; Estimate of difference = 11.88, 95% CI [5.42 to 18.33]
Statistical Analysis 4: Comparison: Ritlecitinib (PF-06651600) 30 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.002922, Miettinen and Nurminen method; Estimate of difference = 9.09, 95% CI [3.10 to 15.07]

3. Secondary Outcome: Percentage of Participants With an Absolute SALT Score of Less Than or Equal to 10 at Week 24: Analysis 1
Description: as for outcome 2
Time Frame: Week 24
Population: FAS included all participants who were randomized, regardless of whether they received study medication. Analysis 1: Participants with missing SALT score at Week 24 due to COVID-19 related reasons excluded from analysis at that time point, participants with missing SALT scores due to other reasons counted as non-responders at that time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo
Number analyzed (Participants) | 124 | 121 | 124 | 119 | 59 | 130
Percentage of participants | 21.77 [14.51 to 29.04] | 13.22 [7.19 to 19.26] | 13.71 [7.66 to 19.76] | 10.92 [5.32 to 16.53] | 1.69 [0.00 to 4.99] | 1.54 [0.00 to 3.65]
Statistical Analysis 1: Comparison: Ritlecitinib (PF-06651600) 200 mg Then 50 mg vs Placebo; Test type: Superiority; p < 0.000001, Miettinen and Nurminen method; Estimate of difference = 20.24, 95% CI [13.23 to 28.49]
Statistical Analysis 2: Comparison: Ritlecitinib (PF-06651600) 200 mg Then 30 mg vs Placebo; Test type: Superiority; p = 0.000337, Miettinen and Nurminen method; Estimate of difference = 11.68, 95% CI [5.82 to 19.07]
Statistical Analysis 3: Comparison: Ritlecitinib (PF-06651600) 50 mg vs Placebo; Test type: Superiority; p = 0.000228, Miettinen and Nurminen method; Estimate of difference = 12.17, 95% CI [6.27 to 19.53]
Statistical Analysis 4: Comparison: Ritlecitinib (PF-06651600) 30 mg vs Placebo; Test type: Superiority; p = 0.001875, Miettinen and Nurminen method; Estimate of difference = 9.39, 95% CI 2-sided [3.86 to 16.46]

4. Secondary Outcome: Percentage of Participants With Patient Global Impression of Change (PGI-C) Score of Moderately Improved or Greatly Improved at Week 24
Description: PGI-C is a self-administered questionnaire to evaluate the improvement or worsening of participant's AA as compared to the start of the study. PGI-C was assessed on a 7-point Likert scale ranged from 1 (greatly improved) to 7 (greatly worsened). Categories were defined based on the PGI-C scores as follows: 1=greatly improved, 2=moderately improved, 3=slightly improved, 4=not changed, 5=slightly worsened, 6=moderately worsened and 7=greatly worsened.
Time Frame: Week 24
Population: FAS included all participants who were randomized, regardless of whether they received study medication. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo
Number analyzed (Participants) | 120 | 119 | 120 | 116 | 55 | 125
Percentage of participants | 52.19 | 45.40 | 49.17 | 41.95 | 11.36 | 9.23
Statistical Analysis 1: Comparison: Ritlecitinib (PF-06651600) 200 mg Then 50 mg vs Placebo; Test type: Superiority; p < 0.000001, Miettinen and Nurminen method; Estimate of difference = 42.96, 95% CI 2-sided [31.68 to 54.25]
Statistical Analysis 2: Comparison: Ritlecitinib (PF-06651600) 200 mg Then 30 mg vs Placebo; Test type: Superiority; p < 0.000001, Miettinen and Nurminen method; Estimate of difference = 36.18, 95% CI 2-sided [25.22 to 47.14]
Statistical Analysis 3: Comparison: Ritlecitinib (PF-06651600) 50 mg vs Placebo; Test type: Superiority; p < 0.000001, Miettinen and Nurminen method; Estimate of difference = 39.96, 95% CI 2-sided [28.85 to 51.06]
Statistical Analysis 4: Comparison: Ritlecitinib (PF-06651600) 30 mg vs Placebo; Test type: Superiority; p < 0.000001, Miettinen and Nurminen method; Estimate of difference = 32.72, 95% CI 2-sided [21.95 to 43.50]

5. Secondary Outcome: Exposure Response of PF-06651600 on Regrowth of Lost Hair Based on Absolute SALT Score of Less Than or Equal to 20 at Week 24: Maximum Effect (Emax) Model
Description: The exposure response of Ritlecitinib (PF-06651600) on the regrowth of scalp hair was characterized using a Bayesian three-parameter hyperbolic Emax model for the SALT score <=20 at Week 24 with an additional term for effect of loading dose. In Emax exposure-response model the response function was the log odds of the percentage of participants with response based on SALT <=20 at Week 24, which was fit on the logistic scale and then back-transformed to percentage. The effect of loading dose is included as fixed factor in the model. The variable that represents loading dose has values of 1 for groups 200/50 mg once daily and 200/30 mg once daily and of 0 for the remaining groups. SALT is a quantitative assessment of AA severity based on the scalp hair loss. The SALT score can vary from 0 (normal) to 100 (severe), with higher scores representing increased severity of disease.
Time Frame: Week 24
Population: FAS included all participants who were randomized, regardless of whether they received study medication. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo
Number analyzed (Participants) | 124 | 121 | 124 | 119 | 59 | 130
Percentage of participants | 32.37 | 20.57 | 22.52 | 13.58 | 4.81 | 1.63

6. Secondary Outcome: Exposure Response of PF-06651600 on Regrowth of Lost Hair Based on Absolute SALT Score of Less Than or Equal to 10 at Week 24: Maximum Effect (Emax) Model
Description: The exposure response of Ritlecitinib (PF-06651600) on the regrowth of scalp hair was characterized using a Bayesian three-parameter hyperbolic Emax model for the SALT score <=10 at Week 24 with an additional term for effect of loading dose. In Emax exposure-response model the response function was the log odds of the percentage of participants with response based on SALT <=10 at Week 24, which was fit on the logistic scale and then back-transformed to percentage. The effect of loading dose is included as fixed factor in the model. The variable that represents loading dose has values of 1 for groups 200/50 mg once daily and 200/30 mg once daily and of 0 for the remaining groups. SALT is a quantitative assessment of AA severity based on the scalp hair loss. The SALT score can vary from 0 (normal) to 100 (severe), with higher scores representing increased severity of disease.
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo
Number analyzed (Participants) | 124 | 121 | 124 | 119 | 59 | 130
Percentage of participants | 21.29 | 13.76 | 14.43 | 9.02 | 3.88 | 1.66

7. Secondary Outcome: Percentage of Participants With an Absolute SALT Score of Less Than or Equal to 20 at Week 4, 8, 12, 18, 28, 34, 40, and 48
Description: SALT is a quantitative assessment of AA severity based on the scalp hair loss. The SALT score can vary from 0 (normal) to 100 (severe), with higher scores representing increased severity of disease.
Time Frame: Week 4, 8, 12, 18, 28, 34, 40, and 48
Population: FAS included all participants who were randomized, regardless of whether they received study medication. Here, "number analyzed" signifies participants evaluable at specific time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Placebo, Ritlecitinib (PF-06651600) 50 mg
Number analyzed (Participants) | 132 | 130 | 130 | 132 | 63 | 65 | 66
Percentage of participants
  Week 4: number analyzed (Participants) | 129 | 124 | 127 | 127 | 62 | 63 | 66
  Week 4 | 0.78 [0.00 to 2.29] | 0.00 [NA to NA] — 95% confidence interval (CI) could not be calculated as there were no participants with SALT score <=20. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=20. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=20. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=20. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=20. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=20.
  Week 8: number analyzed (Participants) | 128 | 121 | 122 | 121 | 62 | 63 | 64
  Week 8 | 5.47 [1.53 to 9.41] | 4.13 [0.59 to 7.68] | 2.46 [0.00 to 5.21] | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=20. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=20. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=20. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=20.
  Week 12: number analyzed (Participants) | 126 | 124 | 126 | 122 | 59 | 61 | 63
  Week 12 | 11.90 [6.25 to 17.56] | 8.87 [3.87 to 13.88] | 6.35 [2.09 to 10.61] | 3.28 [0.12 to 6.44] | 3.39 [0.00 to 8.01] | 1.64 [0.00 to 4.83] | 1.59 [0.00 to 4.67]
  Week 18: number analyzed (Participants) | 121 | 121 | 122 | 117 | 60 | 60 | 62
  Week 18 | 19.83 [12.73 to 26.94] | 13.22 [7.19 to 19.26] | 13.11 [7.12 to 19.10] | 9.40 [4.11 to 14.69] | 3.33 [0.00 to 7.88] | 1.67 [0.00 to 4.91] | 1.61 [0.00 to 4.75]
  Week 28: number analyzed (Participants) | 120 | 119 | 119 | 122 | 60 | 57 | 63
  Week 28 | 34.17 [25.68 to 42.65] | 23.53 [15.91 to 31.15] | 26.05 [18.16 to 33.94] | 20.49 [13.33 to 27.65] | 5.00 [0.00 to 10.51] | 1.75 [0.00 to 5.16] | 6.35 [0.33 to 12.37]
  Week 34: number analyzed (Participants) | 125 | 123 | 124 | 122 | 59 | 61 | 65
  Week 34 | 38.40 [29.87 to 46.93] | 27.64 [19.74 to 35.55] | 33.87 [25.54 to 42.20] | 28.69 [20.66 to 36.71] | 5.08 [0.00 to 10.69] | 19.67 [9.70 to 29.65] | 9.23 [2.19 to 16.27]
  Week 40: number analyzed (Participants) | 128 | 123 | 122 | 120 | 59 | 65 | 65
  Week 40 | 39.06 [30.61 to 47.51] | 33.33 [25.00 to 41.66] | 39.34 [30.68 to 48.01] | 30.00 [21.80 to 38.20] | 6.78 [0.36 to 13.19] | 23.08 [12.83 to 33.32] | 15.38 [6.61 to 24.16]
  Week 48: number analyzed (Participants) | 129 | 122 | 125 | 122 | 61 | 65 | 64
  Week 48 | 39.53 [31.10 to 47.97] | 34.43 [26.00 to 42.86] | 43.20 [34.52 to 51.88] | 31.15 [22.93 to 39.37] | 9.84 [2.36 to 17.31] | 33.85 [22.34 to 45.35] | 18.75 [9.19 to 28.31]

8. Secondary Outcome: Percentage of Participants With an Absolute SALT Score of Less Than or Equal to 10 at Week 4, 8, 12, 18, 28, 34, 40, and 48
Description: SALT is a quantitative assessment of AA severity based on the scalp hair loss. The SALT score can vary from 0 (normal) to 100 (severe), with higher scores representing increased severity of disease. In this outcome measure, percentage of participants with SALT score <=10 were reported.
Time Frame: Week 4, 8, 12, 18, 28, 34, 40, and 48
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Placebo, Ritlecitinib (PF-06651600) 50 mg
Number analyzed (Participants) | 132 | 130 | 130 | 132 | 63 | 65 | 66
Percentage of participants
  Week 4: number analyzed (Participants) | 129 | 124 | 127 | 127 | 62 | 63 | 66
  Week 4 | 0.78 [0.00 to 2.29] | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=10. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=10. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=10. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=10. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=10. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=10.
  Week 8: number analyzed (Participants) | 128 | 121 | 122 | 121 | 62 | 63 | 64
  Week 8 | 2.34 [0.00 to 4.96] | 0.83 [0.00 to 2.44] | 0.82 [0.00 to 2.42] | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=10. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=10. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=10. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=10.
  Week 12: number analyzed (Participants) | 126 | 124 | 126 | 122 | 59 | 61 | 63
  Week 12 | 6.35 [2.09 to 10.61] | 5.65 [1.58 to 9.71] | 5.56 [1.56 to 9.56] | 0.82 [0.00 to 2.42] | 1.69 [0.00 to 4.99] | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with SALT score <=10. | 1.59 [0.00 to 4.67]
  Week 18: number analyzed (Participants) | 121 | 121 | 122 | 117 | 60 | 60 | 62
  Week 18 | 12.40 [6.52 to 18.27] | 7.44 [2.76 to 12.11] | 6.56 [2.16 to 10.95] | 5.13 [1.13 to 9.12] | 1.67 [0.00 to 4.91] | 1.67 [0.00 to 4.91] | 1.61 [0.00 to 4.75]
  Week 28: number analyzed (Participants) | 120 | 119 | 119 | 122 | 60 | 57 | 63
  Week 28 | 29.17 [21.03 to 37.30] | 16.81 [10.09 to 23.53] | 18.49 [11.51 to 25.46] | 16.39 [9.82 to 22.96] | 3.33 [0.00 to 7.88] | 1.75 [0.00 to 5.16] | 3.17 [0.00 to 7.50]
  Week 34: number analyzed (Participants) | 125 | 123 | 124 | 122 | 59 | 61 | 65
  Week 34 | 30.40 [22.34 to 38.46] | 18.70 [11.81 to 25.59] | 23.39 [15.94 to 30.84] | 22.13 [14.76 to 29.50] | 3.39 [0.00 to 8.01] | 13.11 [4.64 to 21.59] | 4.62 [0.00 to 9.72]
  Week 40: number analyzed (Participants) | 128 | 123 | 122 | 120 | 59 | 65 | 65
  Week 40 | 31.25 [23.22 to 39.28] | 25.20 [17.53 to 32.88] | 27.05 [19.17 to 34.93] | 25.00 [17.25 to 32.75] | 3.39 [0.00 to 8.01] | 18.46 [9.03 to 27.89] | 9.23 [2.19 to 16.27]
  Week 48: number analyzed (Participants) | 129 | 122 | 125 | 122 | 61 | 65 | 64
  Week 48 | 33.33 [25.20 to 41.47] | 27.87 [19.91 to 35.82] | 31.20 [23.08 to 39.32] | 25.41 [17.68 to 33.14] | 6.56 [0.35 to 12.77] | 24.62 [14.14 to 35.09] | 14.06 [5.55 to 22.58]

9. Secondary Outcome: Percentage of Participants With at Least 75% Improvement in SALT Score (SALT75) From Baseline at Week 4, 8, 12, 18, 24, 28, 34, 40, and 48
Description: SALT is a quantitative assessment of AA severity based on the scalp hair loss. The SALT score can vary from 0 (normal) to 100 (severe), with higher scores representing increased severity of disease. A SALT 75 response was a 75% or greater reduction from baseline in SALT score.
Time Frame: Week 4, 8, 12, 18, 24, 28, 34, 40, and 48
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Placebo, Ritlecitinib (PF-06651600) 50 mg
Number analyzed (Participants) | 132 | 130 | 130 | 132 | 63 | 65 | 66
Percentage of participants
  Week 4: number analyzed (Participants) | 129 | 124 | 127 | 127 | 62 | 63 | 66
  Week 4 | 0.78 [0.00 to 2.29] | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least 75% improvement in SALT score. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least 75% improvement in SALT score. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least 75% improvement in SALT score. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least 75% improvement in SALT score. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least 75% improvement in SALT score. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least 75% improvement in SALT score.
  Week 8: number analyzed (Participants) | 128 | 121 | 122 | 121 | 62 | 63 | 64
  Week 8 | 4.69 [1.03 to 8.35] | 3.31 [0.12 to 6.49] | 1.64 [0.00 to 3.89] | 0.83 [0.00 to 2.44] | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least 75% improvement in SALT score. | 1.59 [0.00 to 4.67] | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least 75% improvement in SALT score.
  Week 12: number analyzed (Participants) | 126 | 124 | 126 | 122 | 59 | 61 | 63
  Week 12 | 11.90 [6.25 to 17.56] | 8.06 [3.27 to 12.86] | 6.35 [2.09 to 10.61] | 2.46 [0.00 to 5.21] | 1.69 [0.00 to 4.99] | 1.64 [0.00 to 4.83] | 1.59 [0.00 to 4.67]
  Week 18: number analyzed (Participants) | 121 | 121 | 122 | 117 | 60 | 60 | 62
  Week 18 | 20.66 [13.45 to 27.88] | 14.88 [8.54 to 21.22] | 9.84 [4.55 to 15.12] | 11.11 [5.42 to 16.81] | 1.67 [0.00 to 4.91] | 1.67 [0.00 to 4.91] | 1.61 [0.00 to 4.75]
  Week 24: number analyzed (Participants) | 124 | 121 | 124 | 119 | 59 | 65 | 65
  Week 24 | 31.45 [23.28 to 39.62] | 20.66 [13.45 to 27.88] | 22.58 [15.22 to 29.94] | 13.45 [7.32 to 19.57] | 1.69 [0.00 to 4.99] | 1.54 [0.00 to 4.53] | 3.08 [0.00 to 7.28]
  Week 28: number analyzed (Participants) | 120 | 119 | 119 | 122 | 60 | 57 | 63
  Week 28 | 34.17 [25.68 to 42.65] | 24.37 [16.66 to 32.08] | 27.73 [19.69 to 35.77] | 21.31 [14.04 to 28.58] | 5.00 [0.00 to 10.51] | 3.51 [0.00 to 8.29] | 4.76 [0.00 to 10.02]
  Week 34: number analyzed (Participants) | 125 | 123 | 124 | 122 | 59 | 61 | 65
  Week 34 | 38.40 [29.87 to 46.93] | 32.52 [24.24 to 40.80] | 38.71 [30.14 to 47.28] | 28.69 [20.66 to 36.71] | 5.08 [0.00 to 10.69] | 21.31 [11.03 to 31.59] | 10.77 [3.23 to 18.31]
  Week 40: number analyzed (Participants) | 128 | 123 | 122 | 120 | 59 | 65 | 65
  Week 40 | 39.84 [31.36 to 48.33] | 34.96 [26.53 to 43.39] | 42.62 [33.85 to 51.40] | 30.00 [21.80 to 38.20] | 5.08 [0.00 to 10.69] | 23.08 [12.83 to 33.32] | 15.38 [6.61 to 24.16]
  Week 48: number analyzed (Participants) | 129 | 122 | 125 | 122 | 61 | 65 | 64
  Week 48 | 39.53 [31.10 to 47.97] | 36.07 [27.54 to 44.59] | 46.40 [37.66 to 55.14] | 31.15 [22.93 to 39.37] | 9.84 [2.36 to 17.31] | 32.31 [20.94 to 43.68] | 21.88 [11.75 to 32.00]

10. Secondary Outcome: Change From Baseline in SALT Score at Week 4, 8, 12, 18, and 24
Description: SALT is a quantitative assessment of AA severity based on the scalp hair loss. The SALT score can vary from 0 (normal) to 100 (severe), with higher scores representing increased severity of disease. Baseline was defined as pre-dose on Day 1.
Time Frame: Baseline (Day 1), Week 4, 8, 12, 18, and 24
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo
Number analyzed (Participants) | 132 | 130 | 130 | 132 | 63 | 131
Units on a scale
  Change at Week 4: number analyzed (Participants) | 127 | 121 | 124 | 124 | 58 | 127
  Change at Week 4 | -2.3 [-3.64 to -1.01] | -2.7 [-4.03 to -1.35] | -1.8 [-3.16 to -0.50] | -1.3 [-2.60 to 0.06] | -1.3 [-3.19 to 0.69] | -0.9 [-2.17 to 0.46]
  Change at Week 8: number analyzed (Participants) | 124 | 119 | 117 | 115 | 57 | 124
  Change at Week 8 | -12.8 [-15.56 to -10.05] | -12.5 [-15.28 to -9.71] | -6.3 [-9.10 to -3.50] | -5.0 [-7.82 to -2.21] | -1.7 [-5.74 to 2.34] | -1.2 [-3.99 to 1.50]
  Change at Week 12: number analyzed (Participants) | 121 | 120 | 121 | 115 | 56 | 122
  Change at Week 12 | -22.7 [-26.47 to -18.97] | -20.1 [-23.87 to -16.30] | -12.4 [-16.18 to -8.61] | -10.3 [-14.11 to -6.47] | -3.5 [-9.00 to 1.98] | -2.4 [-6.12 to 1.35]
  Change at Week 18: number analyzed (Participants) | 117 | 119 | 117 | 112 | 56 | 119
  Change at Week 18 | -31.2 [-35.63 to -26.83] | -25.0 [-29.41 to -20.55] | -22.5 [-26.94 to -18.07] | -17.5 [-22.02 to -13.02] | -2.4 [-8.87 to 3.97] | -3.9 [-8.31 to 0.43]
  Change at Week 24: number analyzed (Participants) | 118 | 119 | 119 | 114 | 55 | 125
  Change at Week 24 | -36.5 [-41.54 to -31.53] | -29.2 [-34.21 to -24.15] | -33.3 [-38.33 to -28.25] | -23.6 [-28.72 to -18.45] | -4.2 [-11.50 to 3.13] | -5.1 [-10.03 to -0.13]

11. Secondary Outcome: Change From Baseline in SALT Score at Week 28, 34, 40, and 48
Description: as for outcome 10
Time Frame: Baseline (Day 1), Week 28, 34, 40, and 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Placebo, Ritlecitinib (PF-06651600) 50 mg
Number analyzed (Participants) | 132 | 130 | 130 | 132 | 63 | 65 | 66
Units on a scale
  Baseline | 90.3 (15.05) | 90.5 (14.28) | 90.3 (14.69) | 90.0 (15.07) | 88.3 (16.87) | 94.4 (9.31) | 91.5 (13.22)
  Change at Week 28: number analyzed (Participants) | 109 | 113 | 111 | 115 | 55 | 54 | 59
  Change at Week 28 | -44.1 (36.35) | -33.3 (33.85) | -36.1 (33.42) | -29.2 (32.56) | -5.6 (23.15) | -11.5 (22.75) | -5.0 (18.51)
  Change at Week 34: number analyzed (Participants) | 113 | 118 | 117 | 115 | 54 | 59 | 61
  Change at Week 34 | -48.2 (36.16) | -35.5 (35.50) | -43.6 (34.35) | -33.5 (35.01) | -7.6 (23.61) | -27.5 (32.78) | -12.6 (24.47)
  Change at Week 40: number analyzed (Participants) | 116 | 118 | 113 | 109 | 54 | 61 | 60
  Change at Week 40 | -49.3 (36.11) | -38.5 (37.14) | -46.9 (35.68) | -35.9 (35.90) | -11.4 (26.01) | -36.5 (34.56) | -23.0 (30.64)
  Change at Week 48: number analyzed (Participants) | 114 | 112 | 116 | 107 | 53 | 60 | 59
  Change at Week 48 | -49.4 (36.09) | -40.5 (37.27) | -48.9 (36.63) | -40.1 (35.87) | -13.3 (30.13) | -46.3 (35.51) | -32.2 (32.39)

12. Secondary Outcome: Percentage of Participants With at Least a 2 Grade Improvement From Baseline or a Score of 3 in Eyebrow Assessment (EBA) Score (Among Participants Without Normal EBA at Baseline) at Week 4, 8, 12, 18, 24, 28, 34, 40, and 48
Description: EBA is a numeric rating scale developed to characterize eyebrow hair loss. The numeric rating scale ranges from 0 (none) to 3 (normal), where, 0= no eyebrow, 1=minimal eyebrow, 2=moderate eyebrow and 3= normal eyebrow, where higher scores represent less hair loss of eyebrows.
Time Frame: Week 4, 8, 12, 18, 24, 28, 34, 40, and 48
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Placebo, Ritlecitinib (PF-06651600) 50 mg
Number analyzed (Participants) | 132 | 130 | 130 | 132 | 63 | 65 | 66
Percentage of participants
  Week 4: number analyzed (Participants) | 107 | 104 | 104 | 107 | 51 | 53 | 52
  Week 4 | 1.87 [0.00 to 4.44] | 2.88 [0.00 to 6.10] | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least a 2-grade improvement or a score of 3 in EBA. | 0.93 [0.00 to 2.76] | 1.96 [0.00 to 5.77] | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least a 2-grade improvement or a score of 3 in EBA. | 3.85 [0.00 to 9.07]
  Week 8: number analyzed (Participants) | 107 | 101 | 101 | 102 | 52 | 53 | 51
  Week 8 | 10.28 [4.53 to 16.03] | 13.86 [7.12 to 20.60] | 2.97 [0.00 to 6.28] | 4.90 [0.71 to 9.09] | 3.85 [0.00 to 9.07] | 3.77 [0.00 to 8.90] | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least a 2-grade improvement or a score of 3 in EBA.
  Week 12: number analyzed (Participants) | 105 | 103 | 104 | 105 | 48 | 51 | 50
  Week 12 | 22.86 [14.83 to 30.89] | 17.48 [10.14 to 24.81] | 9.62 [3.95 to 15.28] | 7.62 [2.54 to 12.69] | 6.25 [0.00 to 13.10] | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least a 2-grade improvement or a score of 3 in EBA. | 4.00 [0.00 to 9.43]
  Week 18: number analyzed (Participants) | 101 | 101 | 101 | 101 | 49 | 50 | 49
  Week 18 | 29.70 [20.79 to 38.61] | 18.81 [11.19 to 26.43] | 17.82 [10.36 to 25.29] | 12.87 [6.34 to 19.40] | 10.20 [1.73 to 18.68] | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least a 2-grade improvement or a score of 3 in EBA. | 8.16 [0.50 to 15.83]
  Week 24: number analyzed (Participants) | 103 | 102 | 100 | 102 | 48 | 55 | 52
  Week 24 | 33.98 [24.83 to 43.13] | 25.49 [17.03 to 33.95] | 29.00 [20.11 to 37.89] | 16.67 [9.43 to 23.90] | 8.33 [0.51 to 16.15] | 3.64 [0.00 to 8.58] | 5.77 [0.00 to 12.11]
  Week 28: number analyzed (Participants) | 100 | 100 | 99 | 105 | 49 | 48 | 50
  Week 28 | 37.00 [27.54 to 46.46] | 29.00 [20.11 to 37.89] | 27.27 [18.50 to 36.05] | 24.76 [16.51 to 33.02] | 12.24 [3.07 to 21.42] | 4.17 [0.00 to 9.82] | 6.00 [0.00 to 12.58]
  Week 34: number analyzed (Participants) | 104 | 104 | 101 | 105 | 48 | 51 | 52
  Week 34 | 41.35 [31.88 to 50.81] | 30.77 [21.90 to 39.64] | 34.65 [25.37 to 43.93] | 31.43 [22.55 to 40.31] | 14.58 [4.60 to 24.57] | 15.69 [5.71 to 25.67] | 13.46 [4.18 to 22.74]
  Week 40: number analyzed (Participants) | 106 | 102 | 100 | 104 | 50 | 55 | 52
  Week 40 | 43.40 [33.96 to 52.83] | 30.39 [21.47 to 39.32] | 39.00 [29.44 to 48.56] | 33.65 [24.57 to 42.74] | 16.00 [5.84 to 26.16] | 20.00 [9.43 to 30.57] | 26.92 [14.87 to 38.98]
  Week 48: number analyzed (Participants) | 107 | 101 | 101 | 105 | 50 | 55 | 51
  Week 48 | 42.99 [33.61 to 52.37] | 32.67 [23.53 to 41.82] | 43.56 [33.89 to 53.23] | 33.33 [24.32 to 42.35] | 16.00 [5.84 to 26.16] | 30.91 [18.70 to 43.12] | 31.37 [18.64 to 44.11]

13. Secondary Outcome: Percentage of Participants With at Least a 2 Grade Improvement From Baseline or a Score of 3 in Eyelash Assessment (ELA) Score (Among Participants Without Normal ELA at Baseline) at Week 4, 8, 12, 18, 24, 28, 34, 40, and 48
Description: ELA is a numeric rating scale developed to characterize eyelash hair loss. The numeric rating scale ranges from 0 (none) to 3 (normal), where, 0=no eyelash, 1=minimal eyelash, 2=moderate eyelash and 3=normal eyelash, where higher scores represent less hair loss of eyelash.
Time Frame: Week 4, 8, 12, 18, 24, 28, 34, 40, and 48
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Placebo, Ritlecitinib (PF-06651600) 50 mg
Number analyzed (Participants) | 132 | 130 | 130 | 132 | 63 | 65 | 66
Percentage of participants
  Week 4: number analyzed (Participants) | 99 | 93 | 93 | 97 | 44 | 49 | 46
  Week 4 | 3.03 [0.00 to 6.41] | 1.08 [0.00 to 3.17] | 5.38 [0.79 to 9.96] | 1.03 [0.00 to 3.04] | 4.55 [0.00 to 10.70] | 2.04 [0.00 to 6.00] | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least a 2-grade improvement or a score of 3 in ELA.
  Week 8: number analyzed (Participants) | 99 | 90 | 91 | 92 | 45 | 49 | 45
  Week 8 | 9.09 [3.43 to 14.75] | 4.44 [0.19 to 8.70] | 8.79 [2.97 to 14.61] | 4.35 [0.18 to 8.51] | 2.22 [0.00 to 6.53] | 2.04 [0.00 to 6.00] | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least a 2-grade improvement or a score of 3 in ELA.
  Week 12: number analyzed (Participants) | 97 | 91 | 94 | 95 | 42 | 47 | 44
  Week 12 | 16.49 [9.11 to 23.88] | 10.99 [4.56 to 17.41] | 11.70 [5.20 to 18.20] | 7.37 [2.11 to 12.62] | 4.76 [0.00 to 11.20] | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least a 2-grade improvement or a score of 3 in ELA. | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least a 2-grade improvement or a score of 3 in ELA.
  Week 18: number analyzed (Participants) | 94 | 90 | 90 | 91 | 43 | 46 | 43
  Week 18 | 25.53 [16.72 to 34.35] | 20.00 [11.74 to 28.26] | 20.00 [11.74 to 28.26] | 12.09 [5.39 to 18.79] | 6.98 [0.00 to 14.59] | 2.17 [0.00 to 6.39] | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least a 2-grade improvement or a score of 3 in ELA.
  Week 24: number analyzed (Participants) | 96 | 89 | 90 | 92 | 41 | 51 | 46
  Week 24 | 30.21 [21.02 to 39.39] | 21.35 [12.84 to 29.86] | 28.89 [19.52 to 38.25] | 26.09 [17.11 to 35.06] | 4.88 [0.00 to 11.47] | 9.80 [1.64 to 17.97] | 0.00 [NA to NA] — 95% CI could not be calculated as there were no participants with at least a 2-grade improvement or a score of 3 in ELA.
  Week 28: number analyzed (Participants) | 94 | 88 | 87 | 95 | 42 | 44 | 44
  Week 28 | 29.79 [20.54 to 39.03] | 25.00 [15.95 to 34.05] | 36.78 [26.65 to 46.91] | 24.21 [15.60 to 32.82] | 4.76 [0.00 to 11.20] | 6.82 [0.00 to 14.27] | 4.55 [0.00 to 10.70]
  Week 34: number analyzed (Participants) | 97 | 91 | 90 | 95 | 41 | 48 | 46
  Week 34 | 34.02 [24.59 to 43.45] | 26.37 [17.32 to 35.43] | 38.89 [28.82 to 48.96] | 26.32 [17.46 to 35.17] | 7.32 [0.00 to 15.29] | 16.67 [6.12 to 27.21] | 6.52 [0.00 to 13.66]
  Week 40: number analyzed (Participants) | 98 | 89 | 89 | 94 | 43 | 51 | 46
  Week 40 | 39.80 [30.10 to 49.49] | 28.09 [18.75 to 37.43] | 38.20 [28.11 to 48.30] | 27.66 [18.62 to 36.70] | 18.60 [6.97 to 30.24] | 25.49 [13.53 to 37.45] | 17.39 [6.44 to 28.34]
  Week 48: number analyzed (Participants) | 99 | 88 | 90 | 95 | 43 | 51 | 45
  Week 48 | 38.38 [28.80 to 47.96] | 29.55 [20.01 to 39.08] | 40.00 [29.88 to 50.12] | 30.53 [21.27 to 39.79] | 20.93 [8.77 to 33.09] | 37.25 [23.99 to 50.52] | 35.56 [21.57 to 49.54]

14. Secondary Outcome: Percentage of Participants With Patient Global Impression of Change (PGI-C) Score of Moderately Improved or Greatly Improved at Week 4, 8, 12, 18, 24, 34, 40, and 48
Description: as for outcome 4
Time Frame: Week 4, 8, 12, 18, 24, 34, 40, and 48
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Placebo, Ritlecitinib (PF-06651600) 50 mg
Number analyzed (Participants) | 132 | 130 | 130 | 132 | 63 | 65 | 66
Percentage of participants
  Week 4: greatly improved: number analyzed (Participants) | 129 | 124 | 127 | 127 | 62 | 63 | 65
  Week 4: greatly improved | 5.43 | 4.03 | 2.36 | 0 | 0 | 0 | 0
  Week 4: moderately improved: number analyzed (Participants) | 129 | 124 | 127 | 127 | 62 | 63 | 65
  Week 4: moderately improved | 3.10 | 11.29 | 4.72 | 7.87 | 1.61 | 1.59 | 1.54
  Week 8: greatly improved: number analyzed (Participants) | 128 | 121 | 123 | 121 | 61 | 63 | 64
  Week 8: greatly improved | 17.19 | 14.88 | 8.13 | 4.13 | 1.64 | 1.59 | 1.56
  Week 8: moderately improved: number analyzed (Participants) | 128 | 121 | 123 | 121 | 61 | 63 | 64
  Week 8: moderately improved | 13.28 | 21.49 | 7.32 | 16.53 | 4.92 | 3.17 | 4.69
  Week 12: greatly improved: number analyzed (Participants) | 127 | 124 | 125 | 123 | 59 | 60 | 63
  Week 12: greatly improved | 22.83 | 22.58 | 13.60 | 12.20 | 3.39 | 0 | 3.17
  Week 12: moderately improved: number analyzed (Participants) | 127 | 124 | 125 | 123 | 59 | 60 | 63
  Week 12: moderately improved | 18.11 | 19.35 | 14.40 | 14.63 | 3.39 | 10.00 | 7.94
  Week 18: greatly improved: number analyzed (Participants) | 123 | 121 | 122 | 119 | 61 | 60 | 61
  Week 18: greatly improved | 27.64 | 22.31 | 18.03 | 19.33 | 1.64 | 1.67 | 3.28
  Week 18: moderately improved: number analyzed (Participants) | 123 | 121 | 122 | 119 | 61 | 60 | 61
  Week 18: moderately improved | 23.58 | 23.97 | 27.87 | 15.13 | 6.56 | 10.00 | 4.92
  Week 24: greatly improved: number analyzed (Participants) | 126 | 121 | 125 | 121 | 60 | 65 | 65
  Week 24: greatly improved | 36.51 | 26.45 | 28.80 | 28.93 | 1.67 | 1.54 | 4.62
  Week 24: moderately improved: number analyzed (Participants) | 126 | 121 | 125 | 121 | 60 | 65 | 65
  Week 24: moderately improved | 16.67 | 20.66 | 20.80 | 13.22 | 10.00 | 9.23 | 3.08
  Week 34: greatly improved: number analyzed (Participants) | 125 | 121 | 123 | 122 | 59 | 59 | 64
  Week 34: greatly improved | 43.20 | 35.54 | 37.40 | 31.97 | 5.08 | 18.64 | 7.81
  Week 34: moderately improved: number analyzed (Participants) | 125 | 121 | 123 | 122 | 59 | 59 | 64
  Week 34: moderately improved | 12.00 | 17.36 | 15.45 | 15.57 | 6.78 | 22.03 | 20.31
  Week 40: greatly improved: number analyzed (Participants) | 128 | 124 | 122 | 120 | 59 | 65 | 65
  Week 40: greatly improved | 43.75 | 34.68 | 37.70 | 30.00 | 6.78 | 30.77 | 13.85
  Week 40: moderately improved: number analyzed (Participants) | 128 | 124 | 122 | 120 | 59 | 65 | 65
  Week 40: moderately improved | 15.63 | 14.52 | 14.75 | 19.17 | 11.86 | 24.62 | 15.38
  Week 48: greatly improved: number analyzed (Participants) | 129 | 123 | 125 | 122 | 61 | 64 | 64
  Week 48: greatly improved | 44.96 | 33.33 | 42.40 | 31.15 | 6.56 | 42.19 | 26.56
  Week 48: moderately improved: number analyzed (Participants) | 129 | 123 | 125 | 122 | 61 | 64 | 64
  Week 48: moderately improved | 13.18 | 18.70 | 13.60 | 18.03 | 9.84 | 17.19 | 17.19

15. Secondary Outcome: Change From Baseline in Alopecia Areata Patient Priority Outcomes (AAPPO) Domain Scores at Week 4, 8, 12, 18, and 24: Emotional Symptoms and Activity Limitations
Description: AAPPO scale is 11-item self-administered questionnaire that measured hair loss, emotional symptoms, and activity limitations over past week. Items 1-4 assessed current hair loss, eyebrow loss, eyelash loss and body hair loss and were analyzed separately on scale of 0-4, with 0 ='no hair loss' and 4='complete hair loss'. Items 5-8 assessed emotional symptoms. Response choices on these items were scored from 0 ='never' to 4='always'. Items 9-11 assessed activity limitations. Response choices on these items were scored from 0='not at all' to 4='completely'. Change from baseline in AAPPO emotional symptoms sub score were calculated as mean of items 5-8 and ranged from 0(never) to 4(always), where higher scores indicated more emotional symptoms. Change from baseline in AAPPO activity limitations sub score was calculated as mean of items 9-11 and ranged from 0(not at all) to 4(completely), where higher scores indicated more activity limitations. Baseline was defined as pre-dose on Day 1.
Time Frame: Baseline (Day 1), Week 4, 8, 12, 18, and 24
Population: FAS included all participants who were randomized, regardless of whether they received study medication. Here, "number analyzed" signifies participants evaluable at specified time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo
Number analyzed (Participants) | 132 | 130 | 130 | 132 | 63 | 131
Units on a scale
  Change at Week 4: emotional symptoms: number analyzed (Participants) | 127 | 121 | 123 | 122 | 58 | 124
  Change at Week 4: emotional symptoms | -0.37 [-0.49 to -0.25] | -0.22 [-0.34 to -0.10] | -0.33 [-0.45 to -0.21] | -0.31 [-0.44 to -0.19] | -0.29 [-0.47 to -0.11] | -0.28 [-0.40 to -0.16]
  Change at Week 8: emotional symptoms: number analyzed (Participants) | 122 | 119 | 117 | 115 | 56 | 123
  Change at Week 8: emotional symptoms | -0.50 [-0.62 to -0.38] | -0.46 [-0.58 to -0.34] | -0.50 [-0.62 to -0.37] | -0.36 [-0.48 to -0.23] | -0.45 [-0.62 to -0.27] | -0.39 [-0.51 to -0.27]
  Change at Week 12: emotional symptoms: number analyzed (Participants) | 122 | 120 | 119 | 116 | 56 | 121
  Change at Week 12: emotional symptoms | -0.53 [-0.66 to -0.40] | -0.54 [-0.67 to -0.41] | -0.48 [-0.61 to -0.34] | -0.49 [-0.63 to -0.36] | -0.50 [-0.69 to -0.31] | -0.36 [-0.49 to -0.23]
  Change at Week 18: emotional symptoms: number analyzed (Participants) | 118 | 119 | 116 | 114 | 57 | 118
  Change at Week 18: emotional symptoms | -0.64 [-0.78 to -0.51] | -0.57 [-0.71 to -0.44] | -0.60 [-0.74 to -0.46] | -0.54 [-0.68 to -0.40] | -0.44 [-0.63 to -0.24] | -0.43 [-0.56 to -0.29]
  Change at Week 24: emotional symptoms: number analyzed (Participants) | 120 | 118 | 119 | 116 | 55 | 125
  Change at Week 24: emotional symptoms | -0.61 [-0.75 to -0.46] | -0.61 [-0.76 to -0.47] | -0.69 [-0.83 to -0.54] | -0.58 [-0.72 to -0.43] | -0.49 [-0.70 to -0.28] | -0.47 [-0.61 to -0.33]
  Change at Week 4: activity limitations: number analyzed (Participants) | 127 | 121 | 123 | 122 | 58 | 125
  Change at Week 4: activity limitations | -0.19 [-0.29 to -0.08] | -0.04 [-0.15 to 0.07] | -0.16 [-0.27 to -0.05] | -0.13 [-0.24 to -0.02] | -0.20 [-0.36 to -0.04] | -0.18 [-0.29 to -0.07]
  Change at Week 8: activity limitations: number analyzed (Participants) | 122 | 119 | 117 | 115 | 56 | 123
  Change at Week 8: activity limitations | -0.24 [-0.34 to -0.13] | -0.25 [-0.36 to -0.14] | -0.18 [-0.29 to -0.07] | -0.09 [-0.20 to 0.02] | -0.21 [-0.37 to -0.05] | -0.20 [-0.31 to -0.09]
  Change at Week 12: activity limitations: number analyzed (Participants) | 122 | 120 | 119 | 116 | 56 | 121
  Change at Week 12: activity limitations | -0.27 [-0.38 to -0.17] | -0.22 [-0.32 to -0.11] | -0.21 [-0.32 to -0.11] | -0.24 [-0.35 to -0.13] | -0.27 [-0.42 to -0.11] | -0.21 [-0.32 to -0.11]
  Change at Week 18: activity limitations: number analyzed (Participants) | 118 | 119 | 116 | 114 | 57 | 118
  Change at Week 18: activity limitations | -0.35 [-0.45 to -0.24] | -0.26 [-0.36 to -0.15] | -0.23 [-0.34 to -0.12] | -0.23 [-0.34 to -0.12] | -0.28 [-0.44 to -0.13] | -0.26 [-0.36 to -0.15]
  Change at Week 24: activity limitations: number analyzed (Participants) | 120 | 118 | 119 | 115 | 55 | 125
  Change at Week 24: activity limitations | -0.30 [-0.40 to -0.20] | -0.30 [-0.40 to -0.20] | -0.31 [-0.41 to -0.21] | -0.28 [-0.38 to -0.18] | -0.31 [-0.45 to -0.16] | -0.29 [-0.39 to -0.19]

16. Secondary Outcome: Change From Baseline in Alopecia Areata Patient Priority Outcomes (AAPPO) Domain Scores at Week 34, 40, and 48: Emotional Symptoms and Activity Limitations
Description: as for outcome 15
Time Frame: Baseline (Day 1), Week 34, 40, and 48
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Placebo, Ritlecitinib (PF-06651600) 50 mg
Number analyzed (Participants) | 132 | 130 | 130 | 132 | 63 | 65 | 66
Units on a scale
  Change at Week 34: emotional symptoms: number analyzed (Participants) | 112 | 116 | 114 | 113 | 53 | 57 | 60
  Change at Week 34: emotional symptoms | -0.78 (0.95) | -0.72 (1.00) | -0.72 (0.93) | -0.71 (1.06) | -0.62 (0.83) | -0.77 (0.92) | -0.64 (0.91)
  Change at Week 40: emotional symptoms: number analyzed (Participants) | 115 | 119 | 112 | 110 | 54 | 62 | 60
  Change at Week 40: emotional symptoms | -0.84 (1.04) | -0.80 (1.02) | -0.81 (0.98) | -0.83 (1.11) | -0.62 (0.96) | -0.83 (1.01) | -0.66 (1.00)
  Change at Week 48: emotional symptoms: number analyzed (Participants) | 114 | 112 | 115 | 107 | 53 | 60 | 59
  Change at Week 48: emotional symptoms | -0.96 (0.99) | -0.84 (1.07) | -0.85 (1.04) | -0.72 (1.15) | -0.50 (0.89) | -0.98 (1.05) | -0.68 (1.03)
  Change at Week 34: activity limitations: number analyzed (Participants) | 112 | 116 | 114 | 115 | 53 | 57 | 60
  Change at Week 34: activity limitations | -0.37 (0.71) | -0.31 (0.78) | -0.26 (0.73) | -0.37 (0.78) | -0.33 (0.76) | -0.36 (0.59) | -0.42 (0.78)
  Change at Week 40: activity limitations: number analyzed (Participants) | 115 | 119 | 112 | 110 | 54 | 62 | 60
  Change at Week 40: activity limitations | -0.44 (0.76) | -0.33 (0.84) | -0.25 (0.68) | -0.42 (0.81) | -0.23 (0.71) | -0.40 (0.66) | -0.39 (0.84)
  Change at Week 48: activity limitations: number analyzed (Participants) | 114 | 112 | 115 | 107 | 53 | 60 | 59
  Change at Week 48: activity limitations | -0.43 (0.79) | -0.39 (0.84) | -0.29 (0.76) | -0.36 (0.85) | -0.26 (0.90) | -0.44 (0.71) | -0.36 (0.81)

17. Secondary Outcome: Percentage of Participants With Improvement From Baseline on Alopecia Areata Patient Priority Outcomes (AAPPO) Items 1-4 at Week 4, 8, 12, 18, 24, 34, 40, and 48
Description: AAPPO scale is a 11-item self-administered questionnaire that measured hair loss, emotional symptoms, and activity limitations over the past week. Items 1-4 were to assess the current hair loss, eyebrow loss, eyelash loss and body hair loss and were analyzed separately on a scale of 0-4, with 0 ='no hair loss' and 4='complete hair loss', where higher scores indicated more hair loss.
Time Frame: Week 4, 8, 12, 18, 24, 34, 40, and 48
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Placebo, Ritlecitinib (PF-06651600) 50 mg
Number analyzed (Participants) | 132 | 130 | 130 | 132 | 63 | 65 | 66
Percentage of participants
  Week 4: current hair loss on scalp: number analyzed (Participants) | 123 | 123 | 120 | 124 | 59 | 63 | 63
  Week 4: current hair loss on scalp | 11.38 [5.77 to 16.99] | 9.76 [4.51 to 15.00] | 4.17 [0.59 to 7.74] | 4.84 [1.06 to 8.62] | 1.69 [0.00 to 4.99] | 6.35 [0.33 to 12.37] | 3.17 [0.00 to 7.50]
  Week 8: current hair loss on scalp: number analyzed (Participants) | 122 | 120 | 116 | 118 | 58 | 63 | 62
  Week 8: current hair loss on scalp | 11.48 [5.82 to 17.13] | 16.67 [10.00 to 23.33] | 7.76 [2.89 to 12.63] | 8.47 [3.45 to 13.50] | 1.72 [0.00 to 5.07] | 4.76 [0.00 to 10.02] | 8.06 [1.29 to 14.84]
  Week 12: current hair loss on scalp: number analyzed (Participants) | 121 | 123 | 118 | 120 | 56 | 60 | 61
  Week 12: current hair loss on scalp | 20.66 [13.45 to 27.88] | 19.51 [12.51 to 26.52] | 12.71 [6.70 to 18.72] | 13.33 [7.25 to 19.42] | 3.57 [0.00 to 8.43] | 6.67 [0.35 to 12.98] | 4.92 [0.00 to 10.34]
  Week 18: current hair loss on scalp: number analyzed (Participants) | 117 | 120 | 116 | 116 | 58 | 60 | 59
  Week 18: current hair loss on scalp | 27.35 [19.27 to 35.43] | 25.00 [17.25 to 32.75] | 13.79 [7.52 to 20.07] | 16.38 [9.64 to 23.11] | 8.62 [1.40 to 15.84] | 8.33 [1.34 to 15.33] | 6.78 [0.36 to 13.19]
  Week 24: current hair loss on scalp: number analyzed (Participants) | 120 | 120 | 118 | 118 | 57 | 65 | 63
  Week 24: current hair loss on scalp | 35.83 [27.25 to 44.41] | 30.00 [21.80 to 38.20] | 26.27 [18.33 to 34.21] | 24.58 [16.81 to 32.34] | 5.26 [0.00 to 11.06] | 10.77 [3.23 to 18.31] | 6.35 [0.33 to 12.37]
  Week 34: current hair loss on scalp: number analyzed (Participants) | 119 | 119 | 116 | 119 | 56 | 59 | 62
  Week 34: current hair loss on scalp | 42.02 [33.15 to 50.89] | 34.45 [25.92 to 42.99] | 29.31 [21.03 to 37.59] | 30.25 [22.00 to 38.51] | 7.14 [0.40 to 13.89] | 22.03 [11.46 to 32.61] | 11.29 [3.41 to 19.17]
  Week 40: current hair loss on scalp: number analyzed (Participants) | 122 | 123 | 115 | 117 | 56 | 65 | 63
  Week 40: current hair loss on scalp | 41.80 [33.05 to 50.56] | 36.59 [28.07 to 45.10] | 35.65 [26.90 to 44.41] | 32.48 [23.99 to 40.96] | 8.93 [1.46 to 16.40] | 29.23 [18.17 to 40.29] | 19.05 [9.35 to 28.74]
  Week 48: current hair loss on scalp: number analyzed (Participants) | 123 | 122 | 118 | 119 | 58 | 65 | 62
  Week 48: current hair loss on scalp | 42.28 [33.55 to 51.01] | 33.61 [25.22 to 41.99] | 42.37 [33.46 to 51.29] | 32.77 [24.34 to 41.21] | 8.62 [1.40 to 15.84] | 33.85 [22.34 to 45.35] | 20.97 [10.83 to 31.10]
  Week 4: current hair loss on eyebrows: number analyzed (Participants) | 99 | 98 | 94 | 96 | 46 | 48 | 46
  Week 4: current hair loss on eyebrows | 9.09 [3.43 to 14.75] | 7.14 [2.04 to 12.24] | 7.45 [2.14 to 12.75] | 4.17 [0.17 to 8.16] | 4.35 [0.00 to 10.24] | 6.25 [0.00 to 13.10] | 8.70 [0.55 to 16.84]
  Week 8: current hair loss on eyebrows: number analyzed (Participants) | 98 | 95 | 92 | 91 | 46 | 48 | 45
  Week 8: current hair loss on eyebrows | 17.35 [9.85 to 24.84] | 21.05 [12.85 to 29.25] | 11.96 [5.33 to 18.59] | 10.99 [4.56 to 17.41] | 6.52 [0.00 to 13.66] | 4.17 [0.00 to 9.82] | 11.11 [1.93 to 20.29]
  Week 12: current hair loss on eyebrows: number analyzed (Participants) | 97 | 97 | 94 | 94 | 43 | 45 | 44
  Week 12: current hair loss on eyebrows | 27.84 [18.92 to 36.75] | 27.84 [18.92 to 36.75] | 18.09 [10.30 to 25.87] | 15.96 [8.55 to 23.36] | 11.63 [2.05 to 21.21] | 11.11 [1.93 to 20.29] | 6.82 [0.00 to 14.27]
  Week 18: current hair loss on eyebrows: number analyzed (Participants) | 94 | 95 | 91 | 91 | 45 | 45 | 42
  Week 18: current hair loss on eyebrows | 27.66 [18.62 to 36.70] | 33.68 [24.18 to 43.19] | 27.47 [18.30 to 36.64] | 19.78 [11.60 to 27.96] | 13.33 [3.40 to 23.27] | 11.11 [1.93 to 20.29] | 7.14 [0.00 to 14.93]
  Week 24: current hair loss on eyebrows: number analyzed (Participants) | 96 | 94 | 92 | 92 | 44 | 50 | 46
  Week 24: current hair loss on eyebrows | 32.29 [22.94 to 41.65] | 32.98 [23.47 to 42.48] | 30.43 [21.03 to 39.84] | 29.35 [20.04 to 38.65] | 6.82 [0.00 to 14.27] | 12.00 [2.99 to 21.01] | 10.87 [1.87 to 19.86]
  Week 34: current hair loss on eyebrows: number analyzed (Participants) | 96 | 93 | 90 | 94 | 43 | 44 | 45
  Week 34: current hair loss on eyebrows | 42.71 [32.81 to 52.60] | 38.71 [28.81 to 48.61] | 38.89 [28.82 to 48.96] | 31.91 [22.49 to 41.34] | 16.28 [5.24 to 27.31] | 22.73 [10.34 to 35.11] | 13.33 [3.40 to 23.27]
  Week 40: current hair loss on eyebrows: number analyzed (Participants) | 97 | 95 | 90 | 92 | 45 | 50 | 46
  Week 40: current hair loss on eyebrows | 42.27 [32.44 to 52.10] | 36.84 [27.14 to 46.54] | 38.89 [28.82 to 48.96] | 38.04 [28.12 to 47.96] | 20.00 [8.31 to 31.69] | 32.00 [19.07 to 44.93] | 23.91 [11.59 to 36.24]
  Week 48: current hair loss on eyebrows: number analyzed (Participants) | 98 | 94 | 91 | 94 | 45 | 50 | 45
  Week 48: current hair loss on eyebrows | 44.90 [35.05 to 54.75] | 34.04 [24.46 to 43.62] | 43.96 [33.76 to 54.15] | 39.36 [29.49 to 49.24] | 15.56 [4.97 to 26.14] | 38.00 [24.55 to 51.45] | 33.33 [19.56 to 47.11]
  Week 4: current hair loss on eyelashes: number analyzed (Participants) | 87 | 87 | 79 | 86 | 38 | 45 | 38
  Week 4: current hair loss on eyelashes | 11.49 [4.79 to 18.20] | 4.60 [0.20 to 9.00] | 7.59 [1.75 to 13.44] | 9.30 [3.16 to 15.44] | 5.26 [0.00 to 12.36] | 8.89 [0.57 to 17.20] | 5.26 [0.00 to 12.36]
  Week 8: current hair loss on eyelashes: number analyzed (Participants) | 86 | 85 | 78 | 81 | 38 | 45 | 37
  Week 8: current hair loss on eyelashes | 17.44 [9.42 to 25.46] | 17.65 [9.54 to 25.75] | 12.82 [5.40 to 20.24] | 14.81 [7.08 to 22.55] | 7.89 [0.00 to 16.47] | 6.67 [0.00 to 13.95] | 8.11 [0.00 to 16.90]
  Week 12: current hair loss on eyelashes: number analyzed (Participants) | 85 | 86 | 79 | 84 | 36 | 41 | 36
  Week 12: current hair loss on eyelashes | 29.41 [19.73 to 39.10] | 26.74 [17.39 to 36.10] | 16.46 [8.28 to 24.63] | 19.05 [10.65 to 27.44] | 8.33 [0.00 to 17.36] | 14.63 [3.82 to 25.45] | 8.33 [0.00 to 17.36]
  Week 18: current hair loss on eyelashes: number analyzed (Participants) | 83 | 85 | 76 | 81 | 38 | 41 | 34
  Week 18: current hair loss on eyelashes | 31.33 [21.35 to 41.30] | 37.65 [27.35 to 47.95] | 21.05 [11.89 to 30.22] | 22.22 [13.17 to 31.28] | 7.89 [0.00 to 16.47] | 12.20 [2.18 to 22.21] | 2.94 [0.00 to 8.62]
  Week 24: current hair loss on eyelashes: number analyzed (Participants) | 86 | 83 | 77 | 82 | 36 | 46 | 38
  Week 24: current hair loss on eyelashes | 31.40 [21.59 to 41.20] | 42.17 [31.54 to 52.79] | 31.17 [20.82 to 41.51] | 28.05 [18.33 to 37.77] | 8.33 [0.00 to 17.36] | 13.04 [3.31 to 22.78] | 2.63 [0.00 to 7.72]
  Week 34: current hair loss on eyelashes: number analyzed (Participants) | 85 | 82 | 75 | 84 | 35 | 42 | 37
  Week 34: current hair loss on eyelashes | 40.00 [29.59 to 50.41] | 36.59 [26.16 to 47.01] | 37.33 [26.39 to 48.28] | 34.52 [24.36 to 44.69] | 11.43 [0.89 to 21.97] | 21.43 [9.02 to 33.84] | 13.51 [2.50 to 24.53]
  Week 40: current hair loss on eyelashes: number analyzed (Participants) | 86 | 84 | 76 | 82 | 37 | 46 | 38
  Week 40: current hair loss on eyelashes | 43.02 [32.56 to 53.49] | 39.29 [28.84 to 49.73] | 32.89 [22.33 to 43.46] | 36.59 [26.16 to 47.01] | 10.81 [0.81 to 20.82] | 28.26 [15.25 to 41.27] | 13.16 [2.41 to 23.91]
  Week 48: current hair loss on eyelashes: number analyzed (Participants) | 86 | 83 | 76 | 84 | 37 | 46 | 38
  Week 48: current hair loss on eyelashes | 41.86 [31.43 to 52.29] | 37.35 [26.94 to 47.76] | 38.16 [27.24 to 49.08] | 34.52 [24.36 to 44.69] | 8.11 [0.00 to 16.90] | 39.13 [25.03 to 53.23] | 28.95 [14.53 to 43.37]
  Week 4: current hair loss on body: number analyzed (Participants) | 96 | 97 | 96 | 94 | 47 | 47 | 44
  Week 4: current hair loss on body | 11.46 [5.09 to 17.83] | 9.28 [3.50 to 15.05] | 10.42 [4.31 to 16.53] | 6.38 [1.44 to 11.32] | 2.13 [0.00 to 6.25] | 4.26 [0.00 to 10.03] | 11.36 [1.99 to 20.74]
  Week 8: current hair loss on body: number analyzed (Participants) | 95 | 94 | 93 | 89 | 46 | 47 | 43
  Week 8: current hair loss on body | 14.74 [7.61 to 21.86] | 15.96 [8.55 to 23.36] | 13.98 [6.93 to 21.03] | 10.11 [3.85 to 16.38] | 2.17 [0.00 to 6.39] | 6.38 [0.00 to 13.37] | 11.63 [2.05 to 21.21]
  Week 12: current hair loss on body: number analyzed (Participants) | 94 | 94 | 94 | 91 | 45 | 44 | 42
  Week 12: current hair loss on body | 17.02 [9.42 to 24.62] | 19.15 [11.19 to 27.10] | 14.89 [7.70 to 22.09] | 14.29 [7.10 to 21.48] | 4.44 [0.00 to 10.47] | 11.36 [1.99 to 20.74] | 7.14 [0.00 to 14.93]
  Week 18: current hair loss on body: number analyzed (Participants) | 91 | 92 | 93 | 88 | 47 | 44 | 40
  Week 18: current hair loss on body | 19.78 [11.60 to 27.96] | 25.00 [16.15 to 33.85] | 15.05 [7.79 to 22.32] | 15.91 [8.27 to 23.55] | 10.64 [1.82 to 19.45] | 9.09 [0.60 to 17.59] | 7.50 [0.00 to 15.66]
  Week 24: current hair loss on body: number analyzed (Participants) | 93 | 93 | 93 | 90 | 45 | 49 | 44
  Week 24: current hair loss on body | 25.81 [16.91 to 34.70] | 27.96 [18.84 to 37.08] | 20.43 [12.24 to 28.62] | 22.22 [13.63 to 30.81] | 6.67 [0.00 to 13.95] | 16.33 [5.98 to 26.68] | 11.36 [1.99 to 20.74]
  Week 34: current hair loss on body: number analyzed (Participants) | 93 | 92 | 92 | 92 | 44 | 44 | 43
  Week 34: current hair loss on body | 33.33 [23.75 to 42.91] | 33.70 [24.04 to 43.35] | 31.52 [22.03 to 41.02] | 26.09 [17.11 to 35.06] | 11.36 [1.99 to 20.74] | 22.73 [10.34 to 35.11] | 9.30 [0.62 to 17.98]
  Week 40: current hair loss on body: number analyzed (Participants) | 94 | 94 | 91 | 90 | 46 | 49 | 44
  Week 40: current hair loss on body | 35.11 [25.46 to 44.76] | 36.17 [26.46 to 45.88] | 30.77 [21.29 to 40.25] | 25.56 [16.54 to 34.57] | 8.70 [0.55 to 16.84] | 22.45 [10.77 to 34.13] | 11.36 [1.99 to 20.74]
  Week 48: current hair loss on body: number analyzed (Participants) | 95 | 93 | 93 | 92 | 46 | 49 | 44
  Week 48: current hair loss on body | 34.74 [25.16 to 44.31] | 34.41 [24.75 to 44.06] | 36.56 [26.77 to 46.35] | 30.43 [21.03 to 39.84] | 10.87 [1.87 to 19.86] | 34.69 [21.37 to 48.02] | 20.45 [8.54 to 32.37]

18. Other Pre Specified Outcome: Change From Baseline in Depression Subscale Score of Hospital Anxiety and Depression Scale (HADS) at Weeks 4, 8, 12, and 24
Description: HADS is a validated 14-item PRO measure used to assess states of anxiety and depression over the past week. Items were rated on a 4-point severity scale. The HADS produces 2 scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states with established normal score cut-offs. The instrument have been validated for use by adolescents aged 12 and older. Each subscale comprised of 7 items and the participant responds as to how each item applies to him/her over the past week prior to baseline visit, on 4-point response scale. Separate scores were calculated for anxiety and depression with score ranges from 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score range was from 0 to 21 for depression subscale; higher score indicating greater severity of depression symptoms. Baseline was defined as pre-dose on Day 1.
Time Frame: Baseline (Day 1), Week 4, 8, 12, and 24
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo
Number analyzed (Participants) | 132 | 130 | 130 | 132 | 63 | 131
Units on a scale
  Change at Week 4: number analyzed (Participants) | 126 | 120 | 123 | 121 | 58 | 125
  Change at Week 4 | -0.1 [-0.54 to 0.26] | -0.4 [-0.82 to -0.01] | -0.1 [-0.48 to 0.33] | -0.1 [-0.48 to 0.33] | -0.3 [-0.86 to 0.32] | -0.3 [-0.73 to 0.07]
  Change at Week 8: number analyzed (Participants) | 124 | 119 | 118 | 114 | 56 | 124
  Change at Week 8 | -0.5 [-0.89 to -0.06] | -0.3 [-0.71 to 0.12] | -0.2 [-0.58 to 0.26] | 0.2 [-0.25 to 0.59] | -0.2 [-0.79 to 0.43] | -0.3 [-0.73 to 0.10]
  Change at Week 12: number analyzed (Participants) | 121 | 119 | 119 | 114 | 56 | 120
  Change at Week 12 | -0.6 [-1.04 to -0.21] | -0.4 [-0.81 to 0.03] | 0.0 [-0.45 to 0.39] | 0.1 [-0.32 to 0.53] | -0.5 [-1.07 to 0.15] | -0.1 [-0.53 to 0.30]
  Change at Week 24: number analyzed (Participants) | 120 | 118 | 120 | 116 | 56 | 124
  Change at Week 24 | -0.4 [-0.79 to 0.07] | -0.8 [-1.21 to -0.35] | -0.3 [-0.70 to 0.16] | -0.2 [-0.66 to 0.21] | -0.4 [-1.04 to 0.21] | 0.0 [-0.46 to 0.39]

19. Other Pre Specified Outcome: Change From Baseline in Depression Subscale Score of Hospital Anxiety and Depression Scale (HADS) at Week 48
Description: as for outcome 18
Time Frame: Baseline (Day 1), Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Placebo, Ritlecitinib (PF-06651600) 50 mg
Number analyzed (Participants) | 132 | 130 | 130 | 132 | 63 | 65 | 66
Units on a scale
  Baseline: number analyzed (Participants) | 131 | 130 | 130 | 131 | 63 | 65 | 66
  Baseline | 2.7 (2.60) | 3.0 (3.16) | 2.9 (3.00) | 2.8 (2.99) | 2.8 (2.80) | 3.2 (3.36) | 3.3 (3.54)
  Change at Week 48: number analyzed (Participants) | 118 | 118 | 117 | 111 | 55 | 59 | 60
  Change at Week 48 | -0.7 (2.13) | -0.4 (3.15) | -0.3 (2.67) | -0.6 (2.44) | -0.5 (2.53) | -0.9 (3.25) | -0.4 (3.28)

20. Other Pre Specified Outcome: Change From Baseline in Anxiety Subscale Score of Hospital Anxiety and Depression Scale (HADS) at Weeks 4, 8, 12, and 24
Description: HADS is a validated 14-item PRO measure used to assess states of anxiety and depression over the past week. Items were rated on a 4-point severity scale. The HADS produces 2 scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states with established normal score cut-offs. The instrument have been validated for use by adolescents aged 12 and older. Each subscale comprised of 7 items and the participant responds as to how each item applies to him/her over the past week prior to baseline visit, on 4-point response scale. Separate scores were calculated for anxiety and depression with score ranges from 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score range was from 0 to 21 for anxiety subscale; higher score indicating greater severity of anxiety symptoms. Baseline was defined as pre-dose on Day 1.
Time Frame: Baseline (Day 1), Week 4, 8, 12, and 24
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo
Number analyzed (Participants) | 132 | 130 | 130 | 132 | 63 | 131
Units on a scale
  Change at Week 4: number analyzed (Participants) | 125 | 119 | 123 | 121 | 58 | 125
  Change at Week 4 | -0.3 [-0.78 to 0.08] | -0.4 [-0.79 to 0.08] | -0.4 [-0.79 to 0.08] | -0.5 [-0.97 to -0.10] | -0.6 [-1.25 to 0.02] | -0.1 [-0.54 to 0.32]
  Change at Week 8: number analyzed (Participants) | 123 | 119 | 118 | 114 | 56 | 123
  Change at Week 8 | -0.8 [-1.25 to -0.31] | -0.4 [-0.88 to 0.07] | -0.8 [-1.27 to -0.31] | -0.3 [-0.79 to 0.17] | -0.9 [-1.59 to -0.20] | -0.5 [-0.96 to -0.03]
  Change at Week 12: number analyzed (Participants) | 120 | 119 | 119 | 114 | 56 | 121
  Change at Week 12 | -0.7 [-1.22 to -0.28] | -0.9 [-1.40 to -0.46] | -0.7 [-1.22 to -0.27] | -0.3 [-0.77 to 0.19] | -0.9 [-1.55 to -0.17] | -0.4 [-0.84 to 0.09]
  Change at Week 24: number analyzed (Participants) | 119 | 118 | 120 | 115 | 56 | 124
  Change at Week 24 | -0.8 [-1.26 to -0.25] | -0.7 [-1.19 to -0.18] | -0.8 [-1.28 to -0.27] | -0.3 [-0.76 to 0.26] | -1.0 [-1.69 to -0.21] | -0.6 [-1.06 to -0.07]

21. Other Pre Specified Outcome: Change From Baseline in Anxiety Subscale Score of Hospital Anxiety and Depression Scale (HADS) at Week 48
Description: as for outcome 20
Time Frame: Baseline (Day 1), Week 48
Population: FAS included all participants who were randomized, regardless of whether they received study medication. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable at specific time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Placebo, Ritlecitinib (PF-06651600) 50 mg
Number analyzed (Participants) | 130 | 130 | 130 | 131 | 63 | 65 | 66
Units on a scale
  Baseline | 4.6 (3.84) | 4.5 (3.18) | 4.9 (3.31) | 4.3 (3.42) | 5.2 (3.38) | 5.3 (4.20) | 5.3 (3.70)
  Change at Week 48: number analyzed (Participants) | 117 | 118 | 117 | 111 | 55 | 59 | 60
  Change at Week 48 | -1.0 (2.92) | -0.8 (3.10) | -0.8 (3.09) | -0.5 (3.40) | -1.2 (2.89) | -1.3 (3.31) | -0.5 (4.53)

22. Other Pre Specified Outcome: Percentage of Participants With a Baseline Score Indicative of Depression Achieving Normal Depression Subscale Score of HADS at Week 4, 8, 12, 24, and 48
Description: HADS is a validated 14-item PRO measure used to assess states of anxiety and depression over the past week. Items were rated on a 4-point severity scale. The HADS produces 2 scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states with established normal score cut-offs. The instrument have been validated for use by adolescents aged 12 and older. Each subscale comprised of 7 items and the participant responds as to how each item applies to him/her over the past week prior to baseline visit, on 4-point response scale. Separate scores were calculated for anxiety and depression with score ranges from 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score range was from 0 to 21 for depression subscale; higher score indicating greater severity of depression symptoms.
Time Frame: Week 4, 8, 12, 24 and 48
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Placebo, Ritlecitinib (PF-06651600) 50 mg
Number analyzed (Participants) | 7 | 11 | 13 | 14 | 5 | 5 | 10
Percentage of participants
  Week 4: number analyzed (Participants) | 7 | 10 | 13 | 14 | 5 | 5 | 10
  Week 4 | 42.86 [6.20 to 79.52] | 60.00 [29.64 to 90.36] | 53.85 [26.75 to 80.95] | 42.86 [16.93 to 68.78] | 40.00 [0.00 to 82.94] | 60.00 [17.06 to 100.00] | 50.00 [19.01 to 80.99]
  Week 8: number analyzed (Participants) | 6 | 11 | 12 | 12 | 5 | 4 | 10
  Week 8 | 66.67 [28.95 to 100.00] | 45.45 [16.03 to 74.88] | 58.33 [30.44 to 86.23] | 33.33 [6.66 to 60.01] | 20.00 [0.00 to 55.06] | 50.00 [1.00 to 99.00] | 40.00 [9.64 to 70.36]
  Week 12: number analyzed (Participants) | 6 | 11 | 12 | 13 | 5 | 5 | 8
  Week 12 | 50.00 [9.99 to 90.01] | 63.64 [35.21 to 92.06] | 66.67 [39.99 to 93.34] | 30.77 [5.68 to 55.86] | 20.00 [0.00 to 55.06] | 60.00 [17.06 to 100.00] | 62.50 [28.95 to 96.05]
  Week 24: number analyzed (Participants) | 7 | 11 | 12 | 14 | 4 | 4 | 10
  Week 24 | 71.43 [37.96 to 100.00] | 63.64 [35.21 to 92.06] | 41.67 [13.77 to 69.56] | 42.86 [16.93 to 68.78] | 50.00 [1.00 to 99.00] | 50.00 [1.00 to 99.00] | 50.00 [19.01 to 80.99]
  Week 48: number analyzed (Participants) | 6 | 11 | 12 | 13 | 5 | 5 | 10
  Week 48 | 50.00 [9.99 to 90.01] | 63.64 [35.21 to 92.06] | 58.33 [30.44 to 86.23] | 46.15 [19.05 to 73.25] | 80.00 [44.94 to 100.00] | 60.00 [17.06 to 100.00] | 60.00 [29.64 to 90.36]

23. Other Pre Specified Outcome: Percentage of Participants With a Baseline Score Indicative of Anxiety Achieving Normal Anxiety Subscale Score of HADS at Week 4, 8, 12, 24, and 48
Description: HADS is a validated 14-item PRO measure used to assessed states of anxiety and depression over the past week. Items were rated on a 4-point severity scale. The HADS produces 2 scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states with established normal score cut-offs. The instrument have been validated for use by adolescents aged 12 and older. Each subscale comprised of 7 items and the participant responds as to how each item applies to him/her over the past week prior to baseline visit, on 4-point response scale. Separate scores were calculated for anxiety and depression with score ranges from 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score range was from 0 to 21 for anxiety subscale; higher score indicating greater severity of anxiety symptoms.
Time Frame: Week 4, 8, 12, 24 and 48
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Placebo, Ritlecitinib (PF-06651600) 50 mg
Number analyzed (Participants) | 29 | 22 | 26 | 16 | 15 | 19 | 13
Percentage of participants
  Week 4 | 51.72 [33.54 to 69.91] | 45.45 [24.65 to 66.26] | 34.62 [16.33 to 52.90] | 37.50 [13.78 to 61.22] | 40.00 [15.21 to 64.79] | 31.58 [10.68 to 52.48] | 30.77 [5.68 to 55.86]
  Week 8: number analyzed (Participants) | 28 | 20 | 25 | 12 | 14 | 18 | 13
  Week 8 | 46.43 [27.96 to 64.90] | 50.00 [28.09 to 71.91] | 68.00 [49.71 to 86.29] | 41.67 [13.77 to 69.56] | 71.43 [47.76 to 95.09] | 33.33 [11.56 to 55.11] | 46.15 [19.05 to 73.25]
  Week 12: number analyzed (Participants) | 28 | 19 | 26 | 16 | 14 | 19 | 12
  Week 12 | 50.00 [31.48 to 68.52] | 57.89 [35.69 to 80.10] | 38.46 [19.76 to 57.16] | 56.25 [31.94 to 80.56] | 42.86 [16.93 to 68.78] | 47.37 [24.92 to 69.82] | 41.67 [13.77 to 69.56]
  Week 24: number analyzed (Participants) | 27 | 20 | 26 | 15 | 14 | 18 | 13
  Week 24 | 51.85 [33.01 to 70.70] | 65.00 [44.10 to 85.90] | 50.00 [30.78 to 69.22] | 46.67 [21.42 to 71.91] | 57.14 [31.22 to 83.07] | 44.44 [21.49 to 67.40] | 38.46 [12.02 to 64.91]
  Week 48: number analyzed (Participants) | 26 | 18 | 25 | 14 | 13 | 19 | 12
  Week 48 | 53.85 [34.68 to 73.01] | 66.67 [44.89 to 88.44] | 60.00 [40.80 to 79.20] | 50.00 [23.81 to 76.19] | 61.54 [35.09 to 87.98] | 57.89 [35.69 to 80.10] | 58.33 [30.44 to 86.23]

ADVERSE EVENTS:
Time Frame: Baseline up to 5 weeks after last dose of study drug (maximum up to Week 53)
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety analysis set included all participants who received at least 1 dose of study medication.
Arm/Group | Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Ritlecitinib (PF-06651600) 200 mg Then 30 mg | Ritlecitinib (PF-06651600) 50 mg | Ritlecitinib (PF-06651600) 30 mg | Ritlecitinib (PF-06651600) 10 mg | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg | Placebo, Ritlecitinib (PF-06651600) 50 mg
All-Cause Mortality (participants affected / at risk) | 0/131 | 0/129 | 0/130 | 0/132 | 0/62 | 0/65 | 0/66
Serious Adverse Events (participants affected / at risk) | 4/131 | 2/129 | 2/130 | 1/132 | 2/62 | 0/65 | 3/66
Other Adverse Events (participants affected / at risk) | 84/131 | 76/129 | 81/130 | 77/132 | 32/62 | 39/65 | 39/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ritlecitinib (PF-06651600) 200 mg Then 50 mg (N=131) | Ritlecitinib (PF-06651600) 200 mg Then 30 mg (N=129) | Ritlecitinib (PF-06651600) 50 mg (N=130) | Ritlecitinib (PF-06651600) 30 mg (N=132) | Ritlecitinib (PF-06651600) 10 mg (N=62) | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg (N=65) | Placebo, Ritlecitinib (PF-06651600) 50 mg (N=66)
Appendicitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Empyema (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Conversion disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Suicidal behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ritlecitinib (PF-06651600) 200 mg Then 50 mg (N=131) | Ritlecitinib (PF-06651600) 200 mg Then 30 mg (N=129) | Ritlecitinib (PF-06651600) 50 mg (N=130) | Ritlecitinib (PF-06651600) 30 mg (N=132) | Ritlecitinib (PF-06651600) 10 mg (N=62) | Placebo, Ritlecitinib (PF-06651600) 200 mg Then 50 mg (N=65) | Placebo, Ritlecitinib (PF-06651600) 50 mg (N=66)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5 | 5 | 3 | 0 | 4 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 7 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 4 | 12 | 8 | 0 | 4 | 1
Nausea (Gastrointestinal disorders) | 11 | 3 | 3 | 12 | 3 | 8 | 1
Vomiting (Gastrointestinal disorders) | 6 | 7 | 2 | 5 | 1 | 2 | 3
Fatigue (General disorders) | 4 | 6 | 6 | 6 | 4 | 3 | 2
Folliculitis (Infections and infestations) | 11 | 11 | 8 | 5 | 4 | 4 | 4
Influenza (Infections and infestations) | 8 | 1 | 3 | 3 | 3 | 1 | 0
Nasopharyngitis (Infections and infestations) | 19 | 21 | 18 | 21 | 7 | 7 | 4
Upper respiratory tract infection (Infections and infestations) | 18 | 12 | 11 | 16 | 2 | 7 | 6
Urinary tract infection (Infections and infestations) | 11 | 3 | 1 | 5 | 0 | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 2 | 4 | 2 | 2 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 3 | 3 | 5 | 6 | 0 | 1
Dizziness (Nervous system disorders) | 9 | 8 | 4 | 8 | 1 | 0 | 2
Headache (Nervous system disorders) | 17 | 14 | 16 | 24 | 12 | 8 | 8
Insomnia (Psychiatric disorders) | 3 | 0 | 2 | 1 | 1 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 3 | 3 | 0 | 4 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 3 | 4 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 6 | 1 | 0 | 2 | 5
Acne (Skin and subcutaneous tissue disorders) | 6 | 10 | 12 | 12 | 3 | 5 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 7 | 1 | 3 | 1 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 3 | 7 | 1 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 9 | 9 | 7 | 5 | 1 | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT03732807/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT03732807/SAP_001.pdf